#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for Study to elucidate the association of the Renin-angiotensin system and right ventricular function in mechanically ventilated patients |
| <b>Compound Number</b> | : | GSK2586881 |
| <b>Effective Date</b> | : | 30-JUL-2019 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205821.
- The final RAP has been written with the knowledge that the study / project had been terminated early and describes the agreed strategy of only reporting the primary and secondary outcomes.
- This RAP will be provided to the study team members to convey the content of the SAC deliverable.
- This RAP also captures additional clarifications / details to the Critical components version (e.g. clarifies the algorithm for choosing between TTE and TOE results per variable)

#### RAP Author(s):

| Approver | Date | Approval Method |
|--------------------------------------|-------------|---------------------|
| PPD | 12-JUL-2019 | e-mail (archived in |
| Director (Respiratory Biostatistics) | 12-JUL-2019 | Pharma TMF) |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Review Confirmations:**

| Approver | Date | Review<br>Confirmation<br>Method |
|---|---|---|
| Lead Programmer (Development Biostatistics) | 30-JUL-2019 | e-mail (archived in Pharma TMF) |
| PPD (MD) Project Physician Lead (Discovery Medicine Clinical Pharmacology and Experimental Medicine) | 15-JUL-2019 | e-mail (archived in<br>Pharma TMF) |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Director (Respiratory, Clinical Statistics) | 30-JUL-2019 | e-signature<br>(PharmaTMF) |
| Programming Manager (Clinical Programming) | 29-JUL-2019 | e-signature<br>(PharmaTMF) |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTR | ODUCTION | 6 |
| 2. | SLIMI | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | 7 |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | PLAN | NED ANALYSES | 11 |
| | 3.1. | Interim Analyses | |
| | 3.2. | Final Analyses | 11 |
| 4. | | YSIS POPULATIONS | |
| | 4.1. | Protocol Deviations | 13 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS | 1.1 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.1.<br>5.2. | Baseline Definitions | 14 |
| | 5.2.<br>5.3. | Examination of Covariates, Other Strata and Subgroups | |
| | 5.5. | 5.3.1. Covariates and Other Strata | 14 |
| | | 5.3.2. Examination of Subgroups | |
| | 5.4. | Multiple Comparisons and Multiplicity | |
| | 5. <del>4</del> .<br>5.5. | Display order of Echocardiography endpoints (source: SI.CV) | |
| | 5.6. | Other Considerations for Data Analyses and Data Handling | |
| | 0.0. | Conventions | 17 |
| 6. | STUE | OY POPULATION ANALYSES | 18 |
| Ο. | 6.1. | Overview of Planned Study Population Analyses | |
| 7. | PHAF | RMACODYNAMIC AND BIOMARKER ANALYSES | 19 |
| | 7.1. | Primary Pharmacodynamic/Biomarker Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.5. Statistical Analyses / Methods | 20 |
| | | 7.1.5.1. Statistical Methodology Specification | 25 |
| | 7.2. | Secondary Efficacy Analyses | |
| | | 7.2.1. Endpoint / Variables | |
| | | 7.2.2. Summary Measure | 26 |
| | | 7.2.3. Population of Interest | <mark>27</mark> |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events | 27 |
| | | 7.2.5. Statistical Analyses / Methods | 28 |
| | | 7.2.5.1. Supportive Models to the Primary analysis, | |
| | | using other RAS peptides in place of Ang II | 28 |
| | | 7.2.5.2. Combined model of the joint association of Ang | |
| | | II and Ang (1-7) with RV function | 28 |

| | | | | Analysis of disease incidence within the | |
|---|---|---|---|---|---|
| | | | | nechanically ventilated population | |
| | 7.3. | Explorato | ory Efficacy A | Analyses | 32 |
| 8. | CVEEL | | 'CEC | | 22 |
| ο. | 8.1. | | | yses | |
| | 8.2. | | | nd Other Safety Analyses | |
| | 0.2. | Cillical L | aboratory ar | id Other Salety Analyses | 33 |
| 9. | REFE | RENCES | | | 34 |
| J. | | VLIVOLO. | | | |
| 10. | APPE | NDICES | | | 35 |
| | 10.1. | | | Deviation Management and Definitions for | |
| | - | | | | 35 |
| | | 10.1.1. | Exclusions 1 | from Evaluable Population | 35 |
| | 10.2. | | | e of Activities | |
| | | | | fined Schedule of Events | |
| | 10.3. | Appendix | 3: Assessm | nent Windows | 39 |
| | | | | of Assessment Windows for Analyses | |
| | 10.4. | Appendix | 4: Study Ph | nases and Treatment Emergent Adverse | |
| | | Events | | <del>-</del> | 40 |
| | | 10.4.1. | Study Phas | es | 40 |
| | | | | Study Phases for Concomitant Medication | |
| | 10.5. | Appendix | | play Standards & Handling Conventions | |
| | | 10.5.1. | | Process | |
| | | 10.5.2. | | Standards | |
| | 10.6. | | 6: Derived | and Transformed Data | 43 |
| | | 10.6.1. | | | |
| | | 10.6.2. | | lation | |
| | | 10.6.3. | | ynamic / Biomarker | |
| | | 10.6.4. | | Intubation | |
| | | 10.6.5. | Oxygenation | n Index (OI) | 45 |
| | | 10.6.6. | Echocardio | gram (Choosing between TTE and TOE results | |
| | | 40.07 | | ent statistical analyses) | |
| | | 10.6.7. | | Organ Failure Assessment (SOFA) score | |
| | | 10.6.8. | Oxygen Sat | turation | 51 |
| | | 10.6.9. | Calculation | of PaO2 / FiO2 and SpO2 / FiO2n of ARDATA.ALLCVTS | 51 |
| | 10.7. | | | | |
| | 10.7. | 10.7.1. | | g Standards for Missing Data Withdrawals | |
| | | 10.7.1. | | Missing Data | |
| | | 10.7.2. | | Handling of Missing and Partial Dates/Times | |
| | 10.8. | Annendiy | | f Potential Clinical Importance | |
| | 10.0. | | | Values | |
| | | | | values | |
| | 10.9. | | | tions & Trade Marks | |
| | 10.0. | | | ns | |
| | | 10.9.2. | | S | |
| | 10.10 | | | Data Displays | |
| | | | | y Numbering | |
| | | | | ple Shell Referencing | |
| | | | | S | |
| | | | | lation Tables | |

# 2019N413024\_00 205821

#### CONFIDENTIAL

| 10.10.5. | Safety Tables | 73 |
|----------|---------------------------------------------|----|
| 10.10.6. | Pharmacodynamic and Biomarker Tables | 75 |
| | Pharmacodynamic and Biomarker Figures | |
| 10.10.8. | Statistical Modelling Tables | 79 |
| | Statistical Modelling Figures | |
| | .ICH Listings | |
| | .Non-ICH Listings | |
| | x 11: Example Mock Shells for Data Displays | |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 205821.

The study was terminated early and the agreed reporting strategy is to only produce outputs to support the primary and secondary objectives/endpoints. Selected A&R datasets containing the exploratory endpoints may still be produced to enable future access requests and analyses of such endpoints.

Note: All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology, rather than the term "Participant" (although the terms are interchangeable in this RAP document and its associated datasets/outputs).

| Revision Chronology: | | |
|----------------------|-------------|-------------|
| 2016N294782_00 | 26-APR-2017 | Original |
| 2016N294782_01 | 02-JUN-2017 | Amendment 1 |
| 2016N294782_02 | 27-NOV-2017 | Amendment 2 |
| 2016N294782_03 | 27-FEB-2019 | Amendment 3 |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Except for the planned modelling of the Ang II / Ang(1-7) ratio there were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 3 (27-FEB-2019).

The protocol originally stated that the ratio of Ang II / Ang(1-7) would be derived for each participant and formally modelled using the same approach as the primary endpoint. However, the statistical model fitting will not take place. Modelling the ratio does not adequately represent aspects of the underlying biology. For example if a participants Ang II and Ang(1-7) values were both 10 pg/mL and another's were both 10000 pg/mL their derived ratios would be identical (one). Modelling a simple ratio naïvely implies the same significance and biological effect for each participant, even though they are at completely different places on the underlying concentration response curves. The additional approach to jointly analyzing Ang II and Ang (1-7) described in the protocol (and in Section 7.2.5.1) will now be the sole approach to modelling Ang II / Ang(1-7) ratios. Note: The simple summary statistics for the Ang II / Ang(1-7) ratios will still be produced because they capture information about enzyme activity.

Protocol amendment #3 (27-FEB-2019) increases the duration that a participant may be mechanically ventilated, before they are included in the study – from  $\leq$ 24 hours to  $\leq$ 48 hours. This change has been made to assist enrolment of participants into the study, but the sponsor considers that it will not impact the objectives of the study. Informal checks may be made by the study statistician to confirm this assumption (e.g. visual comparisons

of results grouped by protocol version enrolled under). Any such checks would not be formally documented/reported unless a difference was apparent in which case the likely approach would be to perform additional sensitivity analyses with appropriate adjustments to the original output(s) to account for the protocol version.

At the time of writing the Critical Components RAP recruitment was going to commence under Protocol Amendment #1 and switch to amendment #2 as soon as possible. The initial set of subjects enrolled under amendment #1 have a reduced number of endpoints available because amendment #2 added the following endpoints:

| CRF form | Questions / Endpoint |
|---|---|
| Participant<br>Status | Is the patient being managed with extracoporeal membrane oxygenation? |
| | Is the patient being managed with extracorporeal CO2 (ECCO2R) removal? |
| | What is the GI index? |
| LAB ABGS | PH |
| | Base excess |

The critical components RAP indicated sites may re-consent subjects recruited under protocol amendment #1 and enter any new data into the eCRF and suggested an approach for imputing missing data. However, the missing data approach described in the critical components RAP may not be appropriate to the individual subject's circumstances and so the default will now be to leave any data as missing/not applicable. Only 2x subjects were recruited under protocol amendment #1 (PPD and PPD) so the impact of leaving their data missing/not applicable is unlikely to be influential on the outcome, and following the early termination decision these exploratory endpoints are not going to be analyzed further.

# 2.2. Study Objective(s) and Endpoint(s)

Exploratory objectives/endpoints have been included for completeness, but due to the early termination of the study will not be analysed further (unless they naturally form part of an output related to a primary or secondary objective, in which case they may be included on a case by case basis).

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the association between<br>plasma Ang II levels and RV function<br>in mechanically ventilated participants. | <ul> <li>Ang II levels</li> <li>Echocardiographic measures:</li> <li>Ratio of right ventricular to left ventricular end-diastolic area</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | <ul> <li>Paradoxical septal motion</li> <li>Pulmonary arterial systolic pressure (PASP) estimated from transtricuspid pressure and right atrial pressure or inferior vena cava (IVC) diameter (whichever is available)</li> <li>Up to and including Day 3 of observation</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| <ul> <li>To define the incidence of ACP and PCD in mechanically ventilated participants.</li> <li>To evaluate the association between</li> </ul> | <ul> <li>Presence of PCD, ACP (severe PCD) and severe ACP</li> <li>Up to and including Day 3 of observation</li> <li>Ang(1-7) levels</li> </ul> |
| plasma Ang(1-7) levels, Ang II/ Ang(1-7) ratio and RV function in mechanically ventilated participants. | <ul> <li>Ang II/ Ang(1-7) ratio</li> <li>Echocardiographic measures:</li> <li>Ratio of right ventricular to left ventricular end-diastolic area</li> <li>Paradoxical septal motion</li> </ul> |
| | <ul> <li>PASP estimated from transtricuspid pressure and<br/>right atrial pressure or IVC diameter (whichever is<br/>available)</li> <li>Up to and including Day 3 of observation</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the association between plasma Ang II and Ang(1-7) levels and other measures of right ventricular function in mechanically ventilated participants. | <ul> <li>Ang II, Ang(1-7) levels</li> <li>Echocardiographic measures: <ul> <li>Paradoxical septal motion (systolic eccentricity index)</li> <li>Maximal velocity of s wave (tissue Doppler imaging) at the tricuspid annulus</li> <li>Fractional area contraction (end diastolic area minus end systolic area normalised to end diastolic area)</li> <li>Acceleration time of RV ejection flow</li> <li>Mean acceleration of RV ejection flow (maximum velocity/ acceleration time) at end-expiration and end-inspiration</li> <li>Inferior vena cava (IVC) diameter at end-expiration (if available)</li> <li>Respiratory variations of RV velocity time integral (end-expiration minus end-inspiration normalised to end-expiration)</li> <li>Tricuspid annular plane systolic excursion (TAPSE)</li> </ul> </li> <li>Up to and including Day 3 of observation</li> </ul> |
| | Note: "Mean acceleration of RV ejection flow at end expiration" is omitted from the list of exploratory endpoints in the protocol but is collected as part of the study and may be analysed in the same manner as the above exploratory endpoints |
| To evaluate the association between<br>plasma Ang II and Ang(1-7) levels and<br>other measures of cardiac function<br>and pulmonary hemodynamics in<br>mechanically ventilated participants. | <ul> <li>Ang II and Ang(1-7)</li> <li>Central venous pressure (if available)</li> <li>Mean arterial pressure</li> <li>Echocardiographic measures:</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | <ul> <li>Respiratory variations of diameter of superior vena cava</li> <li>Cardiac output (pulsed wave Doppler, left ventricle (LV) outflow track)</li> <li>LV ejection fraction</li> <li>LV Velocity (E') tissue doppler imaging (TDI) of annulus</li> <li>LV early to late ventricular filling velocities (E/A)</li> <li>Up to and including Day 3 of observation</li> </ul> |
| To characterise disease severity by clinical assessment. | <ul> <li>Oxygen saturation (SpO<sub>2</sub>) via pulse oximetry</li> <li>pH of arterial blood gases</li> <li>PaO<sub>2</sub>/FiO<sub>2</sub> ratio</li> <li>PaCO<sub>2</sub></li> <li>Peak and plateau ventilator pressure</li> <li>PEEP</li> <li>Oxygenation index</li> <li>Static respiratory system compliance</li> <li>Mean airway pressure</li> <li>Driving pressure (plateau pressure – total PEEP)</li> <li>Clinical Safety labs</li> <li>Vital Signs</li> <li>Up to and including Day 3 of observation</li> </ul> |
| To characterise levels of organ dysfunction. | Sequential Organ Failure Assessment (SOFA) score Up to and including Day 3 of observation |
| To assess the association of cardiac<br>and inflammatory biomarkers and RV<br>function. | <ul> <li>PCD and ACP status</li> <li>Biomarkers: for example, cardiac biomarkers (B-type natriuretic peptide (BNP)) or inflammatory biomarkers (cytokines such as IL-6, IL-8 and sTNFR1) may be analysed as sample availability allows</li> <li>Up to and including Day 3 of observation</li> </ul> |
| To evaluate the association between<br>additional markers of the RAS system<br>(if samples permit) and<br>primary/secondary or exploratory<br>endpoints. | Markers could include but are not limited to: Ang(1-5) in relation to primary, secondary or exploratory endpoints if sufficient sample is available Up to and including Day 3 of observation |
| To characterize health outcome measures. | <ul> <li>Duration of intubation</li> <li>Length of hospital stay</li> <li>ICU length of stay</li> <li>Ventilator free days</li> <li>In ICU and hospital mortality</li> <li>Up to 28 days after first echocardiogram</li> </ul> |
| To assess lung ventilation and perfusion distribution (in selected site only). | Lung regional ventilation and perfusion with global inhomogeneity (GI) index Up to and including Day 3 of observation |

#### 2.3. Study Design



# 2.4. Statistical Hypotheses / Statistical Analyses

This study is designed to test the hypothesis that an association exists between RAS peptides, primarily plasma Ang II and Ang(1-7) levels, and RV function in mechanically ventilated patients. No formal statistical hypotheses are being tested in this exploratory study.

#### 3. PLANNED ANALYSES

#### 3.1. Interim Analyses

#### Table 1 Interim analyses

None of the planned interim analyses will take place in study 205821 due to the decision to terminate the study early.

The original interim analysis strategy was going to examine data at

- IA1: Approximately 25 evaluable subjects (Note: This was scheduled for Jan 2019 but delayed due to technical issues with the assay for RAS peptides and the study was terminated before the RAS data became available)
- IA2: Approximately 50 evaluable subjects.
- IA3 (Optional): Approximately 100 evaluable subjects

# 3.2. Final Analyses

The final planned analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol (i.e. after the last participant has completed their 28-day follow-up).
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. Protocol deviation reviews have taken place (See Section 4.1)

(Note: as there is no randomisation and no treatment intervention, the usual steps pertaining to unblinding and release of randomisation codes do not apply.)

#### 4. ANALYSIS POPULATIONS

| Population <sup>1</sup> | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who have been screened. | To aid construction<br>of Consort diagram<br>in any publication |
| Enrolled | All participants who had passed screening and who had appropriate informed consent (via any of the processes described in the protocol). | Summary of Subject<br>Status and Reason<br>for Study Withdrawal |
| | | Summary of Study Populations |
| | | Summary of<br>Exclusions from the |

| Population <sup>1</sup> | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | | Safety/Completed/<br>Evaluable<br>Populations |
| Safety | All participants for whom at least one echocardiograph and/or blood sample has been taken, and who did not retrospectively withdraw the consent. | Study population<br>(excl. specific tables<br>mentioned below) |
| | | Safety |
| Evaluable | All participants for whom PASP, RV size ratio, Ang II and Ang(1-7) data have been recorded for at least one study time point, and who did not retrospectively withdraw the consent (and who still had at least one study time point of data remaining after accounting for any prohibited concomitant medications (for example but not limited to renin inhibitors, ARBs or ACE inhibitors) – See Section 10.1.1). | Pharmacodynamic/<br>Biomarker (excl.<br>disease diagnosis<br>status) |
| Evaluable with<br>Prohibited Con<br>Meds | All participants in the Evaluable population plus any participants who were excluded from the Evaluable population because of prohibited concomitant medications (for example but not limited to renin inhibitors, ARBs or ACE inhibitors) | Sensitivity for Primary analysis (conditional on number of prohibited con meds) |
| Completed <sup>2</sup> | All participants for whom PASP, RV size ratio, Ang II, and Ang(1-7) data have been recorded for all three study days. | Disease diagnosis<br>status |
| At Risk | For the purpose of evaluating ACP/PCD and ARDS incidence rates the participants who satisfy 1) PASP and RV size ratio recorded for all three study days (regardless of the Ang II and Ang(1-7) status) and/or 2) databased ACP/PCD and/or ARDS assessment during the study period (even if they do not have three days' worth of study assessments for the above echo outcomes) provided consent is not withdrawn. | Disease diagnosis<br>status |

#### NOTES:

- 1. Please refer to Section 10.10: List of Data Displays which details the population to be used for each display being generated.
- 2. Modifications to the Completed population listed in study protocol to assist with production of summary and incidence rate calculations for ACP/PCD status (include creating a new population "At Risk" to be used with selected incidence rate displays that is independent of the RAS biomarker availability). The remaining completed population is not formally used, but will provide feasibility information (i.e. could we measure items reliably in the "real world" of the ICU)

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the current version of the Protocol Deviation Management Plan.

- 1. Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- 2. This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

No study treatment is being administered in this study. However, GSK's standard SAS macro reporting tools will still assign each participant a set of treatment variables ("No treatment"). There will not be any treatment comparisons. Tables and Figures will only be presented with a single "No Treatment" column unless they are presented by covariate groupings or subgroups as described in Section 5.3 below.

#### 5.2. Baseline Definitions

At present, no analyses involving a change from baseline are planned since there is no treatment intervention. However, for each endpoint the Baseline will be defined as the earliest evaluable timepoint (if a baseline is required).

#### 5.3. Examination of Covariates, Other Strata and Subgroups

#### 5.3.1. Covariates and Other Strata

The set of potential covariates and other strata that may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses are large.

To facilitate flexible model building and analyses a A&R dataset(s) of potential covariate and grouping variables should be constructed (called ARDATA.ALLCVTS). It would be expected to contain three records per participant (Study Day 1, Day 2 and Day 3 values for time-varying covariates), with subject-level covariates repeated across the three records (a flagging variable should also be created to subset the main dataset to extract one record per subject if analyses only involve subject-level covariates); an illustrative example is shown below

| Subject | Visit | SUBJLEV | AGE | SEX | SAPSII | ARDSX | ARDSI |
|---------|-------|---------|-----|-----|--------|-------|-------|
| PPD | Day 1 | 1 | 35 | М | 12 | N | N |
| | Day 2 | 0 | 35 | М | 12 | N | N |
| | Day 3 | 0 | 35 | М | 12 | N | N |
| | Day 1 | 1 | 43 | F | 16 | Υ | N |
| | Day 2 | 0 | 43 | F | 16 | Υ | Υ |
| | Day 3 | 0 | 43 | F | 16 | Υ | Υ |
| | Day 1 | 1 | 54 | M | 7 | N | N |

Guidance for its construction/algorithms are given in Section 10.6.10.

#### 5.3.2. Examination of Subgroups

The following list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered based on items in ARDATA.ALLCVTS.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to producing the final version of the planned output.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup [ARDATA.ALLCVTS Variable] | Categories |
|---|---|
| ARDS Status [ARDSX] | ARDS, No ARDS (diagnosed at any time in the study) |
| Any PCD or ACP [PCDACPX & PCDACPI] | Yes; No (where Yes = Participant had disease state of PCD or ACP) Group can be applied across all study visits [PCDACPX] or to specific days [PCDACPI] |
| No PCD or ACP [NORVDYSX & NORVDYSI] | Yes; No (where Yes = Participant did not have a disease state of PCD or ACP) Group can be applied across all study visits [NORVDYSX] or to |
| | specific days [NORVDYSI] |
| PCD [PCDX & PCDI] | Yes; No (where Yes implies the worst diagnosis received was Moderate PCD across all study visits [PCDX variable] and Yes implies the worst diagnosis received on the corresponding study day was Moderate PCD [PCDI variable]) |
| ACP [ACPX & ACPI] | Yes; No (where Yes implies the worst diagnosis received was Non-<br>severe ACP across all study visits [ACPX variable] and Yes implies the<br>worst diagnosis received on the corresponding study day was Non-<br>severe ACP [ACPI variable]) |
| Severe ACP [SEVACPX & SEVACPI] | Yes; No (where Yes implies the worst diagnosis received was Severe ACP across all study visits [SEVACPX variable] and Yes implies the worst diagnosis received on the corresponding study day was Severe ACP [SEVACPI variable]) |
| ARDS and No PCD or ACP [ARDNOX] | Yes; No (where Yes implies participant received an ARDS diagnosis but never had PCD or ACP at any time in the study) |
| ARDS and PCD [ARDPCDX] | Yes; No (where Yes implies participant received an ARDS diagnosis but the worst case diagnosis was Moderate PCD at any time in the study) |
| ARDS and ACP [ARDACPX] | Yes; No (where Yes implies participant received an ARDS diagnosis but the worst case diagnosis was Non-severe ACP at any time in the study) |
| ARDS and Severe ACP [ARDSACPX] | Yes; No (where Yes implies participant received an ARDS diagnosis and the worst case diagnosis was Severe ACP at any time in the study) |

# 5.4. Multiple Comparisons and Multiplicity

No adjustments for multiplicity will be made.

# 5.5. Display order of Echocardiography endpoints (source: SI.CV)

Whenever multiple Echocardiography endpoints (found in the CV dataset) are required within the same Table/Listing/Figure and the display ordering is not explicitly stated the following display ordering should be apply:

| Priority Order of presentation | CVTSTCD | Description (Note: the actual label/text would be taken from dataset manager at the time of reporting) |
|---|---|---|
| 1 (1st in T/L/F) | AH001CAL | Pulmonary Artery Systolic Pressure |
| NA | AH001 | Pulmonary Artery Systolic Pressure (eCRF) |
| 2 | AK001 | Ratio of RV to LV End-Diastolic Area |
| 3 | AK002 | Paradoxical Septal Motion |
| 4 | AK015 | Have PCD or ACP |
| 5 | AK016 | Severity of PCD or ACP |
| 6 | AK003 | Systolic Eccentricity Index |
| 7 | AK006 | Max Velocity S Wave at Tricuspid Annulus |
| 8 | AK007 | Fractional Area Contraction |
| 9 | AK008 | Acc Time of RV Ejection Flow (Tacc) |
| 10 | TAPSE | Tricuspid Annular Plane Systol Excursion |
| 11 | AK004 | Transtricuspid Pressure Gradient (TPG) |
| 12 | AK009 | Mean Acc of RV Ejection Flow at End Exp |
| 13 | AK010 | Mean Acc of RV Ejec Flow at End Exp-Insp |
| 14 | AK005 | IVC Diameter at End Expiration |
| 15 | AK011 | Respiratory Variations of RV VTI |
| 16 | AK012 | Respiratory Variations of SVC Diameter |
| 17 | CARDOUT | Cardiac Output (CO) |
| 18 | LVEJ | Left Ventricular Ejection Fraction |
| 19 | AK013 | LV Velocity (E') Tissue of Annulus |
| 20 | AK014 | LV Early to Late Filling Velocities |
| 21 | ERATRIAP | Estimated Right Atrial Pressure |
| 22 | AI001 | Measured Right Atrial Pressure |
| 23 | RAP | Right Atrial Pressure |
| 24 | AD003 | Central Venous Pressure (CVP) |
| NA | AH001src | <do display;="" not="" of="" pasp="" source="" to="" track="" used="" variable=""></do> |

Note: Only display AH001CAL but label it using the AH001 label text (this is because the auto derived eCRF value for PASP; supplied as AH001; may not capture all data cases reliably and so will be re-calculated)

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Reporting Standards for Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Enrolled population, unless otherwise specified.

Study population analyses including analyses of participant disposition, protocol deviations, demographic and baseline characteristics, and prior and concomitant medications will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

Note: Local French law prohibits the collection of Race information, so the race/ethnicity variables would be blank in the datasets and displays.

#### 7. PHARMACODYNAMIC AND BIOMARKER ANALYSES

## 7.1. Primary Pharmacodynamic/Biomarker Analyses

#### 7.1.1. Endpoint / Variables

The following variables may be included in the statistical model:

- Independent variable of interest:
  - o Ang II on Study Days 1, 2 and 3 (after any imputations)
- Dependent (bivariate) variable of interest:
  - o PASP on Study Days 1, 2 and 3
  - o RV size ratio on Study Days 1, 2 and 3
- Potential covariates (to be explored, order listed indicates expected importance):
  - o Centre
  - Age at screening
  - o Sex
  - Use of vasopressors on Study Days 1, 2 and 3
  - o PEEP on Study Days 1, 2 and 3
  - o Proning status on Study Days 1, 2 and 3
  - o BMI at screening
  - o Concurrent use of inhaled nitric oxide on Study Days 1, 2 and 3
  - o Mean airway pressure on Study Days 1, 2 and 3
  - o Tidal Volume on Study Days 1, 2 and 3
  - o ECMO on Study Days 1, 2 and 3
  - o ECCO2R on Study Days 1, 2 and 3
  - o SAPS II at screening
  - o PaO2/FiO2 on Study Days 1, 2 and 3

Additionally, the presence/absence of paradoxical septal motion on Study Days 1, 2 and 3 may be assessed on an informal visual basis.

Note: Since the study was terminated early there may not be sufficient information in the collected data to explore covariate analyses and the covariate exploration process may not take place at all.

#### 7.1.2. Summary Measure

The posterior predictive probability of RV dysfunction in a hypothetical individual for a pre-determined "pre-dose" Ang II value,

The posterior predictive probability of RV dysfunction in a hypothetical individual for a pre-determined "post-dose" Ang II value, and

The difference between the above two probabilities.

#### 7.1.3. Population of Interest

The primary pharmacodynamic analyses will be based on the Evaluable population, unless otherwise specified.

#### 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent events which may lead to missing data for all variables (such as death) would not impact the primary analysis since the planned modelling assumes no lag between RAS peptide concentrations and effect on RV dysfunction (i.e. RAS concentrations on day 1 are not used to predict RV dysfunction on day 2 and if death occurs between day 1 and day 2 this will not impact the planned modelling).

Intercurrent events such as taking a non-permitted con med may require exclusion of post medication data if the con med had the potential to confound the true relationship between RAS peptide and RV dysfunction.

Intercurrent events that result in missing data for one or more of the variables required for the primary analysis (e.g. ECHO view not suitable, lost RAS sample) will result in the exclusion of the impacted timepoint as there is not sufficient information to postulate a suitable imputation model.

#### 7.1.5. Statistical Analyses / Methods

The purpose of the primary analysis is to evaluate the association of biomarkers of the Renin Angiotensin System (RAS), specifically Ang II but secondarily Ang(1-7) with measures of RV function (specifically PASP and RV size ratio in the primary model, and also paradoxical septal motion on a more informal visual basis), whilst taking into account any observable variables that may confound the relationship between the two concepts.

RV function will be measured using PASP and RV size ratio. The general principle underlying all the analyses of RV function and RAS peptide biomarkers will be:

- model the joint distribution of PASP and RV size ratio as a function of the RAS
  peptide(s) in question (together with confounding variables also included as
  covariates),
- choose reference values of the RAS peptide(s) in question and estimate a posterior distribution of PASP and RV size ratio for those given values, and
- use the posterior distribution to determine the probability of RV dysfunction (for a future individual participant), defined (following the definition of moderate/severe pulmonary circulatory disease given in Boissier, 2013) as:
  - $\circ$  PASP > 40 mmHg
  - $\circ$  RV size ratio > 0.6

The advantage of this method is that all the information on the continuous scales of PASP and RV size ratio is maintained throughout the modelling process, and that dichotomising

participants into binary categories takes place at the end after the modelling has been done.

In order to evaluate the estimated effect of administering rhACE2 on RV outcomes (via its effect on the RAS peptides), predictions for the probability of RV dysfunction will be calculated for specific, pre-determined values of RAS peptide measurements that represent reasonable estimates for each RAS peptide both before and after dosing with rhACE2 in this patient population. These values will be hereafter referred to as *reference values* (the first reference value, hereafter referred to as the *pre-dose reference* and the second reference value, hereafter referred to as the *post-dose reference* reflect). Note: the terminology "pre-dose" and "post-dose" should not be taken to imply that investigational product is used in this study; these values should be taken as being borrowed from that interventional study. Furthermore, the term "reference values" in this context should not be interpreted as upper or lower limits to the normal range. They represent the best guess available for a patient's typical experience before and after rhACE2 administration.

Initially, the basic model described below would be attempted. If model convergence issues are encountered with that model it is unlikely that more complicated models involving covariates would fit, and covariate exploration may not be attempted. However, if covariate exploration is attempted the addition of covariates would be dependent on a combination of changes in DIC and expert judgement (including the biological rationale for the covariate and/or global structures of other statistical models fitted to comparable data types). To simplify reporting only model outputs from the final selected model would be formally reported (included in the CPSR), but a description / short justification for the selected model would be included in the CPSR.

At the time of writing, the reference values for Ang II (and for completeness Ang(1-7) and Ang(1-5)) were as follows:

| | ANG II (pg/mL) | ANG 1-7 (pg/mL) | ANG 1-5 (pg/mL)<br>Optional endpoint |
|---|---|---|---|
| "Pre-dose" reference value | 30.0 | 2.0 | n/a |
| "Post-dose" reference value | 8.0 | 30.0 | n/a |

An additional sensitivity analysis (to be computed alongside the above) in case the reference study values are discordant with the observed values will use the observed data to determine the references as follows

| Sensitivity | ANG II (pg/mL) | ANG 1-7 (pg/mL) | ANG 1-5 (pg/mL)<br>Optional endpoint |
|---|---|---|---|
| Sensitivity "Predose" reference value | Upper Quartile of<br>Observed ANG II | Lower Quartile of<br>Observed ANG 1-7 | Lower Quartile of<br>Observed ANG 1-5 |
| Sensitivity "Post-dose" reference value | Lower Limit of Quantification | Upper Quartile of Observed ANG 1-7 | Upper Quartile of<br>Observed ANG 1-5 |

The relationship between Ang II (as the explanatory variable) and the joint bivariate distribution of PASP and RV size ratio (the outcome variables) will be analysed using a Bayesian multivariate linear regression model.

The multivariate normal model is specified as follows:

$$\begin{pmatrix} y_{it1} \\ y_{it2} \end{pmatrix} \sim MVNormal \begin{pmatrix} \mu_{it1} \\ \mu_{it2} \end{pmatrix}, \Sigma$$

where  $y_{iij}$  represents the observed value for the *i*th participant, the *t*th time-point and the *j*th outcome (i.e. j = 1 representing PASP and j = 2 representing RV size ratio),  $\mu_{itj}$  represents the expected value for the *i*th participant, *t*th time-point (t = 1,2,3) and the *j*th outcome (j=1 and j=2 as above), and  $\Sigma$  represents a variance-covariance (vcov) matrix for the two outcome variables.

The expected values,  $\mu_{i \in I}$ , are modelled as follows:

$$\mu_{i e j} = \alpha_i + \beta_i x_i + \gamma_{e j} z_{i e}$$

where:

- $\alpha_j$  is the intercept term for the jth outcome (i.e. PASP or RV size),
- $\beta_j$  represents the vector of slope coefficients for all participant-level variables in the model for the *j*th outcome,
- $x_i$  represents the vector of observed participant-level variables values for the ith participant (if applicable initial model structures would not involve such covariates but Age at Screening and Sex would be added first to be consistent with the study protocol),
- $\gamma_{tj}$  represents the matrix of slope coefficients for all timepoint-level variables in the model for the *j*th outcome at time-point t,
- $z_{it}$  represents the matrix of observed time-point-level variables for the *i*th participant at time-point t (e.g. log10- transformed RAS).

The vcov matrix  $\Sigma$  is specified within each study participant, as a Kronecker product of the inter- and intra-marker vcov matrices Sigma and Tigma, respectively:

$$\Sigma = Sigma \otimes Tigma$$

(the notation (8) represent the Kronecker product)

The  $y_{i=1,2}$  inter-marker vcov matrix

$$Sigma = \begin{pmatrix} \sigma_{y_1}^2 & \sigma_{y_1y_2} \\ \sigma_{y_1y_2} & \sigma_{y_2}^2 \end{pmatrix}$$

assumes a constant inter-marker bivariate correlation,  $\rho_{y_1y_2} = \sigma_{y_1y_2} / \sqrt{\sigma_{y_1}^2 \sigma_{y_2}^2}$ , across  $y_{t,j=1,2}$  measured at the same t. The **Sigma** vcov matrix structure, when  $\sigma_{y_2,y_3} = 0$ , implies independence between both markers.

The  $y_{j=1,2}$  inter-marker vcov matrix assumed as

$$Tigma = \begin{pmatrix} 1 & \rho & \rho^2 \\ \rho & 1 & \rho \\ \rho^2 & \rho & 1 \end{pmatrix}$$

implies an intra-marker AR(1) process structure with common correlation parameter  $\rho$ . The dimension of the T is determined by the number of timepoints (t = 1,2,3) the  $y_{i=1,2}$  marker measurements are measured at. Note: Initial simulation work showed an UN (Unstructured) form of vcov for Tigma results in convergence issues due to parameter estimation issues; hence why AR(1) is preferred. A potential drawback to using Kronecker product is that it forces the inter-marker relationship though time to be the same for both response variables; but the Kronecker product requires estimation of fewer parameters (improved chance of model convergence) and recognises the repeated measures (time) structure whilst allowing it to be handled as a nuisance parameter in the final inferences (albeit with the previous caveat).

Given the above assumptions the  $\binom{y_{i+1}}{y_{i+2}}$  vcov structure is derived as follows:

$$\Sigma = Sigma \otimes Tigma =$$

$$\begin{pmatrix} \sigma_{y_1}^2 & \sigma_{y_1y_2} \\ \sigma_{y_1y_2} & \sigma_{y_2}^2 \end{pmatrix} \otimes \begin{pmatrix} 1 & \rho & \rho^2 \\ \rho & 1 & \rho \\ \rho^2 & \rho & 1 \end{pmatrix} = \begin{pmatrix} \sigma_{y_1}^2 * \begin{pmatrix} 1 & \rho & \rho^2 \\ \rho & 1 & \rho \\ \rho^2 & \rho & 1 \end{pmatrix} & \sigma_{y_1y_2}^2 * \begin{pmatrix} 1 & \rho & \rho^2 \\ \rho & 1 & \rho \\ \rho^2 & \rho & 1 \end{pmatrix} \\ \sigma_{y_1y_2} * \begin{pmatrix} 1 & \rho & \rho^2 \\ \rho & 1 & \rho \\ \rho^2 & \rho & 1 \end{pmatrix} & \sigma_{y_2}^2 * \begin{pmatrix} 1 & \rho & \rho^2 \\ \rho & 1 & \rho \\ \rho^2 & \rho & 1 \end{pmatrix}$$

Uninformative prior distributions are assigned for  $\alpha$ ,  $\beta$ ,  $\gamma$ , **Sigma** and **Tigma** as follows:

- For each  $\alpha_j$  outcome variable a normal distribution with mean zero, large variance (e.g. 1E6) would be used as a non-informative prior,
- each element in the vector  $\beta$  is assigned a distribution with the same specifications as for  $\alpha$ ,
- each element in the matrix  $\gamma$  is assigned a distribution with the same specifications as for  $\alpha$  and the elements of  $\beta$ ,
- S, defined as the inverse of Sigma, is assigned an uninformative Wishart prior distribution:  $S\sim Wishart(R,df)$  where:  $R=\begin{pmatrix} 0.01 & 0 \\ 0 & 0.01 \end{pmatrix}$  and df=3.
- The Tigma parameter  $\rho$  is assigned uninformative uniform prior distribution over [-1,1] interval.
- Note: Simulations suggest that the model convergence is improved if the response variables (or more specifically their covariance parameter estimates) are roughly on the same scale (range). Therefore, if required, the response variables may be re-scaled for model fitting, but model inferences/results should be displayed using the original scale of the response variable.
- Note: Simulation work suggests that model convergence may also be sensitive to the software used (due to the complexities of estimating the vcov parameters and the limitations of Gibbs samplers being most efficient when the priors are conjugate to the likelihood of the parameters; once a Kronecker Product vcov is involved the conjugacy is not spotted automatically by most software). The first intent is to use SAS PROC MCMC, but if that does not work then R may be used (e.g. an appropriate package that implements JAGS) and if R fails then Stan may be used. Although a Bayesian implementation of the above model is desired if convergence issues are encountered then SAS PROC MIXED may be used to estimate the required model parameters (it may also as part of the QC checking of the model)
- Note: For IA1 (and IA2 and final analysis, if required) model simplification may occur to improve model convergence (e.g.  $\gamma$  parameter would only contain terms for the RAS peptides and not other time dependent terms such as separate slopes for each visit and endpoint combination).
- The initial model structure would consist of nine parameters, a slope and intercept for the two linear regressions of RAS biomarker level against outcome (PASP or RV Size raio) (four parameters), four parameters of *Sigma*, and one parameter (ρ) for *Tigma*

Estimates for the posterior distributions of coefficients in the model will be obtained using an MCMC simulation running a suitable number of chains for an appropriate number of iterations each to ensure satisfactory convergence of the MCMC sampling algorithm. Nominally, a minimum of 3 chains would be used to produce the Gelman-Rubin diagnostics, though these numbers may be adjusted as necessary and chain

convergence may require separate model runs (e.g. SAS PROC MCMC requires separate model runs to assess the Gelman-Rubin chain convergence (with a zero burn in); but the final MCMC model used for inference requires a non-zero burn in; necessitating separate modelling runs. However, the final model run should utilise one of the sets of starting parameters used in the Gelman-Rubin investigations).

The corresponding secondary pharmacodynamic analyses (using Ang(1-7), and optionally Ang(1-5), in place of Ang II) and a model including Ang II and Ang(1-7) as joint independent variables of interest may be used to support the primary analysis. Details are provided in Section 7.2.

Posterior estimates for the predictive probability of RV dysfunction will be made for the two sets of reference values of Ang II described above (exception is if joint modelling using Ang II and Ang(1-7) is being attempted). If other covariates are included in the final inference model these predictions should be made using the observed mean value for continuous variables and the observed mode value for categorical variables (exception being terms like CENTRE or SEX which would be predict for the average of the corresponding levels). Note: Observed margins may be used if there is a good clinical rationale to do so (assessed on a covariate by covariate basis).

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed

#### 7.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

See above

#### **Model Specification**

See above

#### **Model Checking & Diagnostics**

 "Bayesian Statistics Best Practice at GSK – Clinical Trials using Bayesian Inference" (effective 20-Apr-2017) gives guidance on model checking and diagnostics that would be applicable to the MCMC modelling in this study.

#### **Model Results Presentation**

See above

#### **Subgroup Analyses**

Not planned.

#### **Sensitivity and Supportive Analyses**

- See above. Only the final (chosen) model form would be used to produce the Tables/Listings/Figure outputs supporting the CPSR.
- If the joint modelling strategy fails then an alternative strategy would be to derive the RV

dysfunction status for each participant (using the same criteria) and analyse the collection of derived binary outcomes, accounting for the repeated measures made on each participant (e.g. logistic regression modelling techniques). The final logit model (including any covariates) would be used to determine the probabilities (and differences) for the sets of "pre and post" dose Ang II reference values to be fed into the decision-making criteria. Any such approach wold be documented in the CSR.

### 7.2. Secondary Efficacy Analyses

#### 7.2.1. Endpoint / Variables

The variables to be included in the secondary pharmacodynamic analysis are the same as for the primary pharmacodynamic analysis, with the addition of the following independent variables:

- Ang(1-7) on Study Days 1, 2 and 3
- (Optionally) Ang(1-5) on Study Days 1, 2 and 3 (if the correlation between Ang(1-7) and Ang(1-5) values is not too high otherwise the analysis would not be expected to add additional insights/value)
- Note: The planned modelling using similar techniques to the primary analysis for the Ang II/Ang(1-7) response on Study Days 1, 2 and 3 will not be attempted.

Incidence rates would be assessed across

- i) the entire study (the outcome taking the value of the worst case observed) and
- ii) on an individual visit basis (Note: Screening and Day 1 data would be combined and labelled as Day 1; the worst case outcome used in any combination)

The following rates would be assessed

- Incidence rates of ARDS diagnosis
- Incidence rates of PCD or ACP (any right ventricular dysfunction; regardless of PCD or ACP severity level)
- Incidence rates of PCD (Moderate PCD (not severe enough to qualify as ACP))
- Incidence rates of Non-severe ACP
- Incidence rates Severe ACP

Additionally, the worst case PCD/ACP diagnosis across the study would be combined with the ARDS diagnosis to form the following categories

- ARDS and No PCD or ACP
- o ARDS and PCD
- o ARDS and Non-Severe ACP
- o ARDS and Severe ACP

# 7.2.2. Summary Measure

For the Ang(1-7) and Ang(1-5) endpoints described above:

• The posterior predictive probability of RV dysfunction for pre-determined "pre-dose" Ang II and Ang(1-7) values (or Ang(1-5)),

- The posterior predictive probability of RV dysfunction for pre-determined "post-dose" Ang II and Ang(1-7) values (or Ang(1-5)), and
- The difference between the two (Note: Although the difference will still be computed as Pre-Post for Ang(1-7) and Ang(1-5) negative values would be a favourable outcome).

For the incidence rate variables

- The At Risk population would be used to filter the individuals going into the subsequent analysis dataset
- For rates relating to an individual visit
  - The big N value would not represent distinct participants but instead represents the maximum number of visits in the analysis dataset (derived by counting the number of subject visits where any ARDS or PCD/ACP assessment was made (expecting three visits per subject but may reduce if subjects withdraw/die before day 3))
  - o the little n value would represent the number of completed visits for that item
  - Freq. represents the number of positive occurrences (Subjects with a Yes response)
  - o Rate (%) = 100 \* Freq. / n [little n]
  - o The 95% CI for the rate (%) should be derived using Wilson Score interval with continuity correction methodology
- For rates relating to the entire study
  - The big N value represents the number of participants for whom an ARDS or PCD/ACP assessment was made at any time in the study
  - Freq. represents the number of positive occurrences (Subjects with a Yes response)
  - o Rate (%) = 100 \* Freq. / N [big N]
  - o The 95% CI for the rate (%) should be derived using Wilson Score interval with continuity correction methodology

Any modifications to the above would be described in the CSR.

#### 7.2.3. Population of Interest

The secondary pharmacodynamic analyses will be based on the Evaluable population, unless otherwise specified.

All analyses involving incidence rate endpoints will be based on the At Risk population unless otherwise specified.

# 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

Since there is no investigational product in the study simplistic approaches will be taken to deal with intercurrent events. Any data driven alternative strategies implemented would be described in the CSR.

#### 7.2.5. Statistical Analyses / Methods

The secondary statistical analyses are divided into three subcategories, with the first being variations on the primary analysis: analyses following the same form as the primary analysis but using a different RAS peptide measurement in place of Ang II.

The second subcategory models the joint association of Ang II and Ang(1-7) on RV function (Note: if the observed data ranges do not permit parameter estimation/model convergence of the proposed model then simpler alternative models may not be attempted; but if they are any methodology would be described in the CSR).

The third subcategory of the secondary analyses is an estimate of disease incidence within the mechanically ventilated population.

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 7.2.5.1. Supportive Models to the Primary analysis, using other RAS peptides in place of Ang II

Supportive models to the primary analysis will be conducted following the same methodology as the primary analysis models (see Section 7.1) but with changes as described below.

The first supportive model will include Ang(1-7) as a time-point-level covariate instead of Ang II, and the corresponding reference value from Section 7.1.5.

Note: An optional supportive model would include Ang(1-5) as a time-point-level covariate instead of Ang II, and the corresponding reference value from Section 7.1.5. This model may be attempted if the Ang II and Ang(1-7) modelling does not produce a clear/consistent outcome and/or the observed level of correlation between Ang(1-5) and Ang(1-7) data is deemed likely to result in a different conclusion (*a priori* expectation Ang(1-7) and Ang(1-5) data will be highly correlated, and so any modelling would be expected to produce similar conclusions and duplication would not add value).

# 7.2.5.2. Combined model of the joint association of Ang II and Ang (1-7) with RV function

#### **Endpoint / Variables**

- PASP and RV Size Ratio on Day 1, Day 2 and Day 3 where available
- Time matched concentration of Ang II (Denoted as A in model specification)
- Time matched concentration of Ang (1-7) (Denoted as B in model specification)

#### **Model Specification**

The relationship between Ang II and Ang(1-7) (as joint explanatory variables) and the

joint bivariate distribution of PASP and RV size ratio (the outcome variables) will be analysed using a Bayesian multivariate non-linear regression model.

For simplicity, the repeated measures aspect of the data structure is not being modelled by first intent and Hill coefficients are assumed to be 1. If data permit, a similar strategy to the primary analysis that accounts for repeated measures may be attempted (e.g. Kronecker product with an AR(1) structure for Tigma), but only the model used for final inference would be reported. If data do not permit the planned model to be fitted no further modelling is proposed. However, if alternative model(s) are attempted and successful, they would be described in the CSR).

The multivariate normal model is specified as follows (for maximum flexibility time has been left in the parameter definitions):

$$\binom{y_{it1}}{y_{it2}} \sim MVNormal \left( \binom{\mu_{it1}}{\mu_{it2}}, \Sigma \right)$$

where  $y_{iij}$  represents the observed value for the *i*th participant, the *t*th time-point and the *j*th outcome (i.e. j = 1 representing PASP and j = 2 representing RV size ratio),  $\mu_{iej}$  represents the expected value for the *i*th participant, *t*th time-point (t = 1,2,3) and the *j*th outcome (t = 1,2,3) and t = 1,2,3 and the *j*th outcome (t = 1,2,3) and t = 1,2,3 and t = 1,2,3 are the two outcome variables.

The expected values,  $\mu_{i \in I}$ , are modelled as follows:

$$= \frac{B asal_{j} + M ax_{Bj} \frac{[B]}{EC_{S0jB|A=0}} + M ax_{Aj} \frac{[A]}{EC_{S0jA|B=0}} + M ax_{ABj} \frac{[A][B]}{EC_{S0jA|B=0} EC_{S0jB|A\to\infty}}}{1 + \frac{[B]}{EC_{S0jB|A=0}} + \frac{[A]}{EC_{S0jA|B=0}} + \frac{[A][B]}{EC_{S0jA|B=0} EC_{S0jB|A\to\infty}}}$$

Where,

Basal<sub>i</sub> is the response in the absence of A and B for the jth outcome

Max<sub>Aj</sub> is the response to saturating concentrations of A in the absence of B for the jth outcome

 $Max_{Bj}$  is the response to saturating concentrations of B in the absence of A for the jth outcome

Max<sub>ABj</sub> is the response in the presence of saturating concentrations of both ligands for the jth outcome

EC<sub>50jA|B=0</sub> is the EC<sub>50</sub> of A in the absence of B for the jth outcome

EC<sub>50iBlA=0</sub> is the EC<sub>50</sub> of B in the absence of A for the jth outcome

 $EC_{50jB|A\to\infty}$  is the  $EC_{50}$  of B in the presence of saturating concentrations of A for the jth outcome

[A] is time matched concentration of AngII (to aid review  $[A_{it}]$  notation not used)

[B] is time matched concentration of Ang(1-7) (to aid review  $[B_{it}]$  notation not used)

Also note that  $EC_{50jA|B=0}$  x  $EC_{50jB|A\to\infty} = EC_{50jB|A=0}$  x  $EC_{50jA|B\to\infty}$ , so the equation is symmetrical in A & B.

The vcov structure for  $\Sigma_{(6x6)}$  is constructed using the same approach as the primary analysis model but with an Identity matrix used for Tigma by first intent

$$\Sigma = Sigma \otimes Tigma =$$

$$\begin{aligned} & \begin{pmatrix} \sigma_{y_1}^2 & \sigma_{y_2,y_2} \\ \sigma_{y_2,y_2} & \sigma_{y_2}^2 \end{pmatrix} \otimes \begin{pmatrix} 1 & 0 & 0 \\ 0 & 1 & 0 \\ 0 & 0 & 1 \end{pmatrix} and \\ & Var \begin{pmatrix} y_{i11} \\ y_{i21} \\ y_{i31} \\ y_{i12} \\ y_{i22} \\ y_{i32} \end{pmatrix} = \begin{pmatrix} \begin{pmatrix} \sigma_{y_1}^2 & 0 & 0 \\ 0 & \sigma_{y_2}^2 & 0 \\ 0 & 0 & \sigma_{y_1}^2 \end{pmatrix} & \begin{pmatrix} \sigma_{y_1,y_2}^2 & 0 & 0 \\ 0 & \sigma_{y_2,y_2}^2 & 0 \\ 0 & \sigma_{y_2,y_2}^2 & 0 & 0 \\ 0 & \sigma_{y_2,y_2}^2 & 0 & 0 \\ 0 & \sigma_{y_2,y_2}^2 & 0 & 0 \\ 0 & \sigma_{y_2,y_2}^2 & 0 & 0 \\ 0 & \sigma_{y_2,y_2}^2 & 0 & 0 \end{pmatrix} \\ & \begin{pmatrix} \sigma_{y_2,y_2}^2 & 0 & 0 \\ 0 & \sigma_{y_2}^2 & 0 & 0 \\ 0 & \sigma_{y_2}^2 & 0 & 0 \\ 0 & 0 & \sigma_{y_2}^2 \end{pmatrix} \end{pmatrix}$$

Uninformative prior distributions are assigned for the parameters as follows:

- Model parameters Basal<sub>j</sub>, Max<sub>Aj</sub>, Max<sub>Bj</sub>, Max<sub>ABj</sub>, EC<sub>50jA|B=0</sub>, EC<sub>50jB|A=0</sub> and EC<sub>50jB|A→∞</sub> (for j=1 (PASP) and 2 (RV Size ratio)) will each be assigned a prior of Normal(Mean=0, Var=1^E6). Note: By first intent these are all independent prior statements and correlation structures between related parameters would be expected to be observed in the observed posterior covariances of the model parameters (see Sensitivity analyses sections for alternative prior structures if model convergence issues are encountered).
- S, defined as the inverse of Sigma, is assigned an uninformative Wishart prior distribution:  $S \sim Wishart(R, df)$  where:  $R = \begin{pmatrix} 0.01 & 0 \\ 0 & 0.01 \end{pmatrix}$  and df = 3.

#### **Model Checking & Diagnostics**

As per Primary analysis

#### **Model Results Presentation**

 Once the model parameters have been estimated analogous predictions of the Posterior Probability of RV dysfunction (and differences between pre and post dose AnglI levels) would be obtained as per Primary analysis. However, twice the number of items would be produced because there would be a need to condition on the two "pre and post dose" values for Ang(1-7) for each set of Ang II values.

#### **Subgroup Analyses**

Not planned

#### **Sensitivity and Supportive Analyses**

- If model convergence issues are encountered the prior structure may be modified to group related sets of parameters together using a MVN (multivariate normal distribution). Two MVN priors distributions may be set up (one for each j) using parameters Basal<sub>j</sub>, Max<sub>Aj</sub>, Max<sub>Bj</sub>, Max<sub>ABj</sub>, EC<sub>50jA|B=0</sub>, EC<sub>50jB|A=0</sub> and EC<sub>50jB|A→∞</sub>. The MVN mean would be a vector of zeros and the prior for the vcov matrix of the model parameters would be an inverse-wishart with R=Identity (7x7) and df=7.
- An AR(1) structure may be attempted for the Tigma vcov matrix and would use an uninformative uniform prior distribution over -1,1 interval for parameter ρ

# 7.2.5.3. Analysis of disease incidence within the mechanically ventilated population

The incidence of ACP and PCD in the population will be presented as summary tables, by study day, and overall (i.e. diagnosis at any time during the three-day study period).

Descriptive statistics (N (population), #Occurrences (Freq.), number at risk (n), Incidence Rate and 95% CI for Rate (methodology for 95% CI: Wilson Score interval with continuity correction))

# 7.3. Exploratory Efficacy Analyses

No exploratory analyses are planned due to the early termination of the study.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 8.1. Adverse Events Analyses

Only Serious Adverse Events (SAEs) relating to study procedures or any GSK medications are being recorded and reported in this study. SAEs will be presented as a summary table and a listing, and will be based on GSK Core Data Standards.

# 8.2. Clinical Laboratory and Other Safety Analyses

Chemistry and Haematology Laboratory evaluations and Vital Signs test results will be presented as summary tables and listings. Additionally, all values of potential clinical importance will be presented as listings, together with all other measurements of the same test in the same participant. These displays will be based on GSK Core Data Standards.

#### 9. REFERENCES

Boissier F, Katsahian S, Razazi K, Thille AW, Roche-Campo F, Leon R, et al. Prevalence and prognosis of cor pulmonale during protective ventilation for acute respiratory distress syndrome. Intensive Care Med. 2013 Oct;39(10):1725-1733.

El-Khatib MF, Jamaleddine GW, A New Oxygenation Index for Reflecting Intrapulmonary Shunting in Patients Undergoing Open-Heart Surgery CHEST 2004; 125:592–596

de Man, Tu, Handoko, et al Dysregulated Renin–Angiotensin–Aldosterone System Contributes to Pulmonary Arterial Hypertension Am J Respir Crit Care Med Vol 186, Iss. 8, pp 780–789, Oct 15, 2012.

Vincent J-L., Moreno R., Takala J., Willatts S., De Mendonca A., Bruning H., Reinhart C.K., Suter P.M., Thijs L.G., The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. Intensive Care Med (1996) 22:707-710

## 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Evaluable Population

## 10.1.1. Exclusions from Evaluable Population

Subjects with major/important protocol deviations will be considered for exclusion from Evaluable Population. The Protocol Deviation Management Plan (PDMP) will be used to determine major/important protocol deviations that will lead to exclusion from the Evaluable Population (Note: In the event the PDMP retains the template text / default terminology which refers to "per protocol population" it would be interpreted as the "Evaluable population" for study 205821).

In addition, a subject meeting any of the following criteria will be excluded from the Evaluable population (or if more applicable, only the relevant timepoint(s) excluded):

| Number | Exclusion Description |
|---|---|
| 01 | Participants whose day 1, day 2 and day 3 samples were all lost or for whom the post sample processing was unable to produce evaluable results would be excluded from the evaluable population If a single day (or two days) are impacted by the above reason(s) then the participant shall remain in the evaluable population, but the impacted time points would be removed from the analysis. |
| 02 | If a single day (or two days) are impacted by the ECHO results that are later deemed of insufficient quality (e.g. this may be discovered by independent review/adjudication of source notes) then those data points would be removed from the analysis (but the participant would remain in the evaluable population). If all of the day 1, day 2 and day 3 ECHO results are impacted in this way then the participant would be removed from the evaluable population. |
| 03 | If the participant takes a prohibited concomitant medication that, in the opinion of the GSK medical monitor, may confound / interfere with the estimation of the true relationship between RAS peptides and an endpoint then any post con-med observations would be removed from the corresponding analysis. |

# 10.2. Appendix 2: Schedule of Activities

# 10.2.1. Protocol Defined Schedule of Events

| Procedure | Study Period | | | Notes | | |
|---|---|---|---|---|---|---|
| | Screening <sup>1</sup> | Day<br>1 | Day<br>2 | Day<br>3 | Up to day<br>28 | |
| Start of mechanical ventilation | Х | | | | | |
| Inclusion/exclusion criteria | Х | | | | | Reason for intubation (underlying diagnosis e.g. sepsis, pneumonia) to be collected where possible. |
| Informed consent (ICF) | Х | | | | | Consent process will be followed as outlined in Informed Consent Process (Section 12.3.3) |
| Demography | Х | | | | | If it is not possible to collect at screening can be collected at any point during the study. |
| Height and weight | Х | | | | | Collected for the purposes of evaluating BMI. Clinical estimates are acceptable if direct measurement is not possible. |
| Medical history | х | | | | | If possible to collect, includes medication and cardiovascular risk factors. If it is not possible to collect at screening can be collected at any point during the study. |
| Diagnosis of<br>pulmonary<br>circulatory<br>dysfunction (PCD)<br>and acute cor<br>pulmonale (ACP) | | Х | Х | Х | | As per echocardiographic output. |
| Participant status | Х | х | х | х | | Intubation status, proned status; diagnosis of acute respiratory distress syndrome (ARDS) including severity at time of diagnosis (if available). Post screening status to be assessed at the same time point as echocardiogram (± 1 hour). |
| Participant<br>management | X | Х | Х | Х | | Management with extracorporeal membrane oxygenation (ECMO) and extracorporeal CO <sub>2</sub> (ECCO <sub>2</sub> R) removal. Post screening status to be assessed at the same time point as echocardiogram (± 1 hour). |
| Procedure | Study Period | | | Notes | | |
|---|---|---|---|---|---|---|
| | Screening <sup>1</sup> | Day<br>1 | Day<br>2 | Day<br>3 | Up to day<br>28 | |
| Simplified acute physiology score (SAPS II) | Х | | | | | To be taken at time of intubation. |
| Sequential Organ<br>Failure (SOFA) score | Х | Х | Х | Х | | |
| Echocardiogram | | X | X | X | | Transthoracic echocardiogram (TTE) and/or transoesophageal echocardiogram (TOE). First echocardiogram must be completed within 48 hours of starting mechanical ventilation (but ≤24 hours, whenever possible); the following echocardiograms will be undertaken as per standard of care 24 hours apart (± 2 hours) on subsequent consecutive days (Day 2 and 3). |
| Vital signs | X <sup>3</sup> | Х | Х | х | | Blood pressure (mean arterial, systolic and diastolic), heart rate, body temperature to match echocardiogram time points (± 30 minutes)². |
| Laboratory assessments | Х | Х | Х | Х | | Clinical chemistry and haematology. |
| Ventilator settings | X <sup>3</sup> | х | х | х | | Includes tidal volume, respiratory rates, static respiratory compliance, level of positive end expiratory pressure (PEEP), peak and plateau ventilator pressures, mean airway pressure and driving pressure. Measurements to be taken at intubation and at the time of each echocardiogram (± 30 mins)². |
| Lung function and blood gas measures | X <sup>3</sup> | X | X | X | | Oxygen saturation (SaO <sub>2</sub> ) via pulse oximetry. Arterial Blood Gases (ABGs) measuring partial pressure of oxygen and carbon dioxide (PaO <sub>2</sub> and PaCO <sub>2</sub> ). <sup>4</sup> Oxygen requirement (FiO <sub>2</sub> ) should be documented at the <u>same</u> time point. pH, lactate and bicarbonate levels and base excess or deficit when available should also be documented when ABGs are assessed. Measurements to be taken at intubation and at the time of each echocardiogram (± 30 mins) <sup>2</sup> . |

| Procedure | | Study Period | | | Notes | |
|---|---|---|---|---|---|---|
| | Screening <sup>1</sup> | Day<br>1 | Day<br>2 | Day<br>3 | Up to day<br>28 | |
| Electrical Impedance<br>Tomography | Х | Х | Х | Х | | Measurements to be taken at intubation and at the time of each echocardiogram when available (±2 hours)². |
| Serious Adverse<br>Event (SAE) Review | <====== | =====> | | | | SAEs will only be collected during the 3 day observation period or until participant withdrawal, whichever is sooner. |
| Concomitant medication review | <====== | :====>> | | | Only specified prescription medication (name, start and end dates required) as described in Section 7.1 of the protocol. Vasopressor use to be documented for each time point of echocardiography. | |
| Intensive Care Unit (ICU) length of stay | | <==: | | | ======> | Will be recorded daily up to 28 days. |
| Ventilator free days | | <==: | ===== | | =====> | Will be recorded daily up to 28 days; however, follow up is not necessary beyond hospital discharge. |
| In hospital mortality | | <==: | ===== | ===== | =====> | Will be recorded daily up to 28 days; however, follow up is not necessary beyond hospital discharge. |
| Biomarkers | Biomarkers | | | | | |
| Blood sample for<br>renin-angiotensin<br>system (RAS)<br>biomarkers | | x x x | | | Blood samples to be taken at the same time as echocardiography (± 30 mins) <sup>2</sup> . | |
| Blood sample for biomarkers | | x x x | | | Blood samples to be taken at the same time as echocardiography (± 30 mins) <sup>2</sup> . | |

- 1. Screening may be considered part of Day 1.
- 2. When multiple measurements are to be taken at the same time in relation to echocardiography, blood sampling for RAS peptides should be given priority. Other measurements (e.g. ventilator settings) to be prioritized as per investigator for patient care.
- 3. Will be recorded at the time of intubation if available.
- 4. Where available, a blood sample is required for arterial blood gases (ABGs) for PaO<sub>2</sub>/FiO<sub>2</sub> and oxygenation index. A FiO<sub>2</sub> measurement should be assessed at the same time point as ABGs are taken for PaO<sub>2</sub>.

# 10.3. Appendix 3: Assessment Windows

# 10.3.1. Definitions of Assessment Windows for Analyses

Data management will maintain the allowable visit/sampling windows for study procedures. Calendar days will be used rather than 24 hour intervals from the start of the 1<sup>st</sup> echo measurement on Day 1, since it is unlikely study procedures will cross midnight. Both date and times are typically collected on the eCRF so if required elapsed times can be used.

# 10.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 10.4.1. Study Phases

## 10.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 4 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

# 10.5.1. Reporting Process

| Software | |
|---|---|
| <ul> <li>The currently supported versions of SAS software will be used. If required, the currently supported<br/>versions of R and STAN software may be used.</li> </ul> | |
| Reporting Area | |
| HARP Server | : UK1SALX00175 |
| HARP Compound | : GSK2586881 |
| Analysis Datasets | Analysis Datasets |
| Analysis datasets | Analysis datasets will be created according to Legacy GSK A&R dataset standards. |
| Generation of RTF Files | |
| RTF files will be g | enerated for the final reporting effort. |

#### 10.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All
  participant level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

#### **Unscheduled Visits**

- Unscheduled will not be included in summary tables and/or figures.
  - If unscheduled visits are included (decision on a case by case basis), the most appropriate method would be used (e.g. summaries displayed by slotting the unscheduled visits to analysis time points

| All unscheduled vis | <ul> <li>as per Section 10.3.1)).</li> <li>All unscheduled visits will be included in listings and figures (when they relate to individual participants <ul> <li>e.g. participant level response vs time profiles).</li> </ul> </li> </ul> |
|---|---|
| <b>Descriptive Summary</b> | Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| <b>Graphical Displays</b> | Graphical Displays |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |
| | se the same plotting symbol/linestyle/colour combination for a participant in all facilitate easy cross comparison across different data types |

#### 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 10.3.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Echo Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Echo Date → Study Day = Ref Date First Echo Date
  - Ref Data ≥ First Echo Date → Study Day = Ref Date (First Echo Date) + 1

#### Study Date/Time (Time 0h)

- Calculated as the elapsed time since the date and time of the first echocardiogram
- Used to align observations of different domains within an individual participant
- Preference to derive using the same algorithm as the HARP standard helper macros and to display
  using an appropriate format to the range of values being displayed (e.g. xx days yy hours zz minutes or
  xx minutes and zz seconds)

•

# 10.6.2. Study Population

#### Age

- Age is approximated as only year of birth is captured:
  - Age = Calendar Year at Time of Informed Consent Year of Birth
  - Age is sometimes referred to in this RAP as Age at Screening (but should be interpreted as Age at time of informed consent)

# 10.6.3. Pharmacodynamic / Biomarker

#### **RAS Biomarkers**

- Ang II/Ang(1-7) is calculated as the ratio of the value of Ang II to the corresponding (same-day) value of Ang(1-7). If either Ang II or Ang(1-7) is missing for a given Study Day then the ratio will also be derived as missing.
- If required Ang II / Ang(1-5) (or any other ratio combination of the RAS peptides) would be derived and processed in an analogous way to the Ang II / Ang(1-7) ratio.

For the derivation of Angll / Ang(1-7) ratios, the following will apply:

| Flag | S | Numerator (ANGII) | | | |
|---|---|---|---|---|---|
| | | BLQ | Data | ALQ | Missing |
| (ANG1-7) | BLQ | (1/2 LLQ of ANGII) /<br>(1/2 LLQ of Ang(1-7)) | ANGII /<br>(1/2 LLQ of Ang(1-<br>7)) | (ULQ of ANGII) /<br>(1/2 LLQ of Ang(1-7)) | Missing |
| | Data | (1/2 LLQ of ANGII) /<br>Ang(1-7) | ANGII / Ang(1-7) | (ULQ of ANGII) /<br>Ang(1-7) | Missing |
| Denominator | ALQ | (1/2 LLQ of ANGII) /<br>(ULQ of Ang(1-7)) | ANGII /<br>(ULQ of Ang(1-7)) | (ULQ of ANGII) /<br>(ULQ of Ang(1-7)) | Missing |
| | Missing Missing | | Missing | Missing | Missing |
| LLQ | / ULQ = Lov | ver / Upper Limit of Quantificat | tion. BLQ / ALQ = Below / | Above Limit of Quantificati | on |

LLQ / ULQ - Lower / Opper Limit of Quantification, BLQ / ALQ - Below / Above Limit of Quantification

Note: The status of the numerator and denominator / outcome should be sufficiently tracked to allow subsequent Summary Tables to display the amount of imputation necessary.

Note: all other pharmacodynamic/biomarker endpoints derived from other items should be auto-calculated on the eCRF and therefore supplied in SI datasets.

In general, it is assumed that biomarker endpoints will require variance stabilising transformations, such as taking a loge transformation prior to analysis (and that summary statistics appropriate to loge normally distributed data will apply for all summaries; log base 10 may also be used in place of natural logarithms). However, this assumption will be considered for each endpoint individually prior to the generation of summary tables or statistical analysis, and if deemed more appropriate, a loge transformation will not be applied, or non-parametric methods may be employed.

If transformations are used then the results will be reported on the back-transformed scale unless otherwise stated.

Unless otherwise specified the following applies to the biomarkers

- Values below LLQ will be set as LLQ/2
- Values above the upper limit of quantification (ULQ) will be set as ULQ
- Imputed values will be used for the purposes of the computation of change from baseline and for summaries, plots and analysis, if deemed applicable.
- Number of data imputed will be highlighted in the summary tables & listings will report the values as below LLQ or above ULQ, alongside the imputed result used in statistical analyses.
- If multiple LLQ's and ULQ's are available per assay (i.e. multiple runs with different standard curves are
  utilised) then the LLQ and/or ULQ value used for the above purposes shall be the minimum of the
  available LLQs and/or the maximum of the BLQ's.

#### 10.6.4. Reason for Intubation

The reason for intubation is captured in the eCRF using a free text field. To allow these items to be summarised succinctly each free text entry will be mapped to a common set of nomenclature. Upon receiving the data transfer associated with the planned data review (e.g. planned interim and/or end of study reporting) a list of the unique free text

entries from the reason for intubation field will be supplied to the medical monitor, who will assign each entry into one of the following categories (Note: each participant may only be assigned to a single category). Additional categories may be added based upon the observed data if deemed necessary by the medical monitor. Only categories that have terms mapped to them need to be displayed. A listing of unique free text terms and the mappings should also be produced (using similar design concepts to the Adverse Event shell AE2)

| ID Number | Allowable mapping of free text |
|-----------|------------------------------------|
| | (display in the order listed here) |
| 0 | Not Applicable (not intubated) |
| 1 | Sepsis |
| 2 | Pneumonia |
| 3 | Acute Respiratory Failure |
| 4 | Cardiac Cause |
| 5 | Neurologic event |
| 6 | Other reason for intubation |
| 7 | No reason for intubation supplied |

# 10.6.5. Oxygenation Index (OI)

The derivation of Oxygenation Index was omitted from the protocol in error and has been documented in the RAP for completeness.

Oxygenation index (OI) (sometimes termed oxygenation factor) is another measure of gas exchange and pulmonary efficiency which factors in the mean airway pressure (Paw) term in the calculation step [El-Khatib, 2004].

It is calculated using Equation 1,

#### Equation 1 Oxygenation index

Oxygenatio n Index (%) = 
$$\frac{\text{FiO2 * Mean Airway Pressure}}{\text{PaO2}}$$
 where Mean Airway Pressure and PaO2 are measured in mmHg and FiO2 is entered as a % and not a proportion

# 10.6.6. Echocardiogram (Choosing between TTE and TOE results for subsequent statistical analyses)

This section describes how to choose which result to select for subsequent statistical analyses when multiple options exist. They are based on the echocardiogram parameters after InForm Post Go Live 3.1 (implemented approx. Jan 2019). Table 2, Table 3, Table 4, Table 5, Table 6 and Table 7 enumerate the possible data combinations and which values to select for the planned echocardiogram endpoints.

Table 2 Selection algorithm (conditional on eCRF input) for the endpoints listed in Table 3

| ID# | eCRF state for TTE<br>(Transthoratic<br>echocardiography) | eCRF state for<br>TOE<br>(Transesophageal<br>echocardiography) | Selected value<br>for statistical<br>analyses | Text value to display in listings |
|---|---|---|---|---|
| 1 | <blank></blank> | <blank></blank> | Missing (".") | No result |
| 2 | <blank></blank> | Not Done | Missing (".") | No result |
| 3 | <blank></blank> | Numerical entry | <toe value=""></toe> | <toe value=""></toe> |
| 4 | Not Done | <blank></blank> | Missing (".") | No result |
| 5 | Not Done | Not Done | Missing (".") | No result |
| 6 | Not Done | Numerical entry | <toe value=""></toe> | <toe value=""></toe> |
| 7 | Numerical entry | <blank></blank> | <tte value=""></tte> | <tte value=""></tte> |
| 8 | Numerical entry | Not Done | <tte value=""></tte> | <tte value=""></tte> |
| 9 | Numerical entry | Numerical entry | <tte value=""></tte> | <tte value=""></tte> |

Table 3 Endpoints to apply the Table 2 selection criteria to

| CVTSTCD | Description |
|---------|------------------------------------------|
| AK001 | Ratio of RV to LV End-Diastolic Area |
| AK003 | Systolic Eccentricity Index |
| AK006 | Max Velocity S Wave at Tricuspid Annulus |
| AK007 | Fractional Area Contraction |
| AK008 | Acc Time of RV Ejection Flow (Tacc) |
| AK009 | Mean Acc of RV Ejection Flow at End Exp |
| AK010 | Mean Acc of RV Ejec Flow at End Exp-Insp |
| AK005 | IVC Diameter at End Expiration |
| AK011 | Respiratory Variations of RV VTI |
| TAPSE | Tricuspid Annular Plane Systol Excursion |
| AK012 | Respiratory Variations of SVC Diameter |
| CARDOUT | Cardiac Output (CO) |
| LVEJ | Left Ventricular Ejection Fraction |
| AK013 | LV Velocity (E') Tissue of Annulus |
| AK014 | LV Early to Late Filling Velocities |

Table 4 Selection algorithm for Paradoxical Septal Motion (CVTSTCD = AK002)

| ID# | eCRF state for TTE<br>(Transthoratic<br>echocardiography) | eCRF state for<br>TOE<br>(Transesophageal<br>echocardiography) | Selected value<br>for statistical<br>analyses | Text value to display in listings |
|---|---|---|---|---|
| 1 | ZZND (Not Done) | ZZND (Not Done) | Missing<br>(" <blank>")</blank> | Not Done |
| 2 | ZZND (Not Done) | N (No) | N | No |
| 3 | ZZND (Not Done) | Y (Yes) | Υ | Yes |
| 4 | N (No) | ZZND (Not Done) | N | No |
| 5 | N (No) | N (No) | N | No |
| 6 | N (No) | Y (Yes) | Υ | Yes |
| 7 | Y (Yes) | ZZND (Not Done) | Υ | Yes |
| 8 | Y (Yes) | N (No) | Υ | Yes |
| 9 | Y (Yes) | Y (Yes) | Y | Yes |

Note: If only one result is present (e.g. a TTE value only but no TOE value databased) then the selected text should be the value present (i.e. Yes, No or Not Done as appropriate to the available result).

Table 5 Selection algorithm for TPG (Trans-tricuspid pressure gradient, CVTSTCD = AK004)

| ID# | eCRF state for TTE<br>(Transthoratic<br>echocardiography) | eCRF state for<br>TOE<br>(Transesophageal<br>echocardiography) | Selected value<br>for statistical<br>analyses | Text value to display in listings |
|---|---|---|---|---|
| 1 | <blank></blank> | <blank></blank> | Missing (".") | No result |
| 2 | <blank></blank> | Numerical entry | <toe value=""></toe> | <toe value=""></toe> |
| 3 | Numerical entry | <blank></blank> | <tte value=""></tte> | <tte value=""></tte> |
| 4 | Numerical entry | Numerical entry | <tte value=""></tte> | <tte value=""></tte> |

Table 6 Selection algorithm for RAP (Right atrial pressure; Potential results could come from either ERATRIAP or Al001 CVTSTCD record but only possible to receive one of those codes for each participant/timepoint combination)

| RAP "Estimated" or "Measured" | ID# | eCRF state<br>for<br>Measured<br>(CVP) | eCRF state for TTE<br>(Transthoratic<br>echocardiography) | eCRF state for TOE<br>(Transesophageal<br>echocardiography) | Selected<br>value for<br>statistical<br>analyses | Text value<br>to display in<br>listings |
|---|---|---|---|---|---|---|
| "Estimated"<br>(i.e. only | 1 | NI/A /NIa | <blank></blank> | <blank></blank> | Missing<br>(".") | No result |
| ÈRATRIAP record | 2 | N/A (No<br>Al001 | <blank></blank> | Numerical entry | <toe<br>value&gt;</toe<br> | <toe<br>value&gt;</toe<br> |
| exists for that | 3 | record) | Numerical entry | <blank></blank> | <tte<br>value&gt;</tte<br> | <tte<br>value&gt;</tte<br> |

| RAP "Estimated" or "Measured" | ID# | eCRF state<br>for<br>Measured<br>(CVP) | eCRF state for TTE<br>(Transthoratic<br>echocardiography) | eCRF state for TOE<br>(Transesophageal<br>echocardiography) | Selected value for statistical analyses | Text value<br>to display in<br>listings |
|---|---|---|---|---|---|---|
| participant / timepoint) | 4 | | Numerical entry | Numerical entry | <tte<br>value&gt;</tte<br> | <tte value=""></tte> |
| "Measured"<br>(i.e. only | 5 | <blank></blank> | | | Missing<br>(".") | No result |
| Al001<br>record<br>exists for<br>that<br>participant /<br>timepoint) | 6 | Numerical<br>entry | N/A (No<br>ERATRIAP<br>record) | N/A (No<br>ERATRIAP<br>record) | <measured value=""></measured> | <measured value=""></measured> |

Note: In the listing of Echocardiogram endpoints when the RAP is "measured" then the TTE and TOE columns should be populated with Not applicable and only the "Selected" column would be populated.

Table 7 Selection algorithm for PASP (Pulmonary artery systolic pressure, CVTSTCD = AH001CAL)

| ID# | Selected TPG value (see Table 5) | Selected RAP value (See Table 6) | Selected value for statistical analyses | Text value to display in listings |
|---|---|---|---|---|
| 1 | Missing (".") | Missing (".") | Missing (".") | No result |
| 2 | Missing (".") | Numerical entry | Missing (".") | No result |
| 3 | Numerical entry | Missing (".") | Missing (".") | No result |
| 4 | Numerical entry | Numerical entry | <tpg +="" rap=""></tpg> | <tgp +="" rap=""></tgp> |

Note: All PASP values in analysis and reporting datasets and consequent tables, listings and figures will be re-derived by stats and programming using the algorithms in Table 7.

PASP values are also automatically derived within the eCRF form and are supplied in the data management transfer of the CV dataset under the CVTSTCD of "AH001". However, it has been noted in test data transfers that the auto calculation does not always derive correct results due to the complexities of the data source combinations (e.g. Participant PPD Day 1 had a TPG from the TOE method but an estimated RAP from the TTE method but the eCRF autocalculation incorrectly supplied a missing PASP value). Therefore there is a need to programmatically re-drive PASP and as a consequence there will be additional records in ARDATA versions of the CV dataset compared to the SI version (CVTSTCD = AH001CAL).

To facilitate sensitivity analyses regarding the frequency/reason of "missing" PASP values an additional variable may be created in ARDATA datasets (as required) that tracks the inputs to the PASP calculation (see Table 8). This tracking variable would not need to be displayed in the listing of echocardiogram endpoints.

Table 8 Additional variable/result to track the derived PASP inputs (assigned a CVTSTCD = AH001src)

| AH001src<br>value | TPG source used in derivation of PASP (see Table 5) | RAP source used in derivation of PASP (See Table 6) |
|---|---|---|
| 1 | Missing (".") | Missing (".") |
| 2 | Missing (".") | TTE |
| 3 | Missing (".") | TOE |
| 4 | Missing (".") | Measured |
| 5 | TTE | Missing (".") |
| 6 | TTE | TTE |
| 7 | TTE | TOE |
| 8 | TTE | Measured |
| 9 | TOE | Missing (".") |
| 10 | TOE | TTE |
| 11 | TOE | TOE |
| 12 | TOE | Measured |

# 10.6.7. Sequential Organ Failure Assessment (SOFA) score

The score will be calculated on a daily basis. Adrenergic agents that do not appear in Vincent, 1996 and for which a highest dose has been recorded, will be assigned a SOFA score of 2. Zero points are assigned if none of the points scoring criteria are met. If any of the information required to derive an individual SOFA component score is missing or cannot be obtained, then that component score will be set to a missing value. The SOFA score will be calculated by summing the individual component scores (individual components derived as below). Note: Central Nervous System component will not be used in deriving the SOFA score in Study 205821:

| | T _ | Т. | Т | | |
|---|---|---|---|---|---|
| SOFA Score /<br>Variable (x) | 0 | 1 | 2 | 3 | 4 |
| Respiration:<br>P <sub>a</sub> O <sub>2</sub> /F <sub>i</sub> O <sub>2</sub><br>(mmHG) | x ≥ 400 | 300 ≤ x < 400 | 200 ≤ x < 300 | $100 \le x < 200$ With Respiratory sup (Note: if $P_aO_2/F_iO_2$ in but subject not on rethen a score of 2 sho | these categories spiratory support |
| Coagulation:<br>Platelets (10^3<br>/ mm^3) | x ≥ 150 | 100 ≤ x<br>< 150 | 50 ≤ x < 100 | 20 ≤ x < 50 | x < 20 |
| Liver:<br>Bilirubin<br>(µmol/L) | x < 20 | 20 ≤ x <<br>33 | $33 \le x < 102$ | 102 ≤ x < 204 | x ≥ 204 |
| Cardiovascular: Hypotension (Adrenergic agents administered for at least one hour; doses are in µg/kg/min) | Mean<br>Arterial<br>Pressur<br>e ≥ 70<br>mmHg | Mean<br>Arterial<br>Pressur<br>e < 70<br>mmHg | Dopamine≤5.<br>0<br>(µg/kg/min)<br>or any dose<br>of:<br>Dobutamine<br>Or any dose<br>of an<br>adrenergic<br>agent not<br>listed here or<br>in Vincent<br>(1996) | Dopamine 5.1-15.0 (µg/kg/min) or Epinephrine≤0.1 or Norepinephrine≤0.1 | Dopamine > 15.0 (µg/kg/min) or Epinephrine>0.1 or Norepinephrine>0.1 |
| Central Nervous System: Glasgow Coma Score | x ≥ 15 | 13 ≤ x ≤<br>14 | 10 ≤ x ≤ 12 | $6 \le x \le 9$ | x < 6 |
| Renal:<br>Creatinine<br>(μmol/L) | x ≤ 110 | 110 < x<br>≤ 170 | 170 < x ≤ 300 | 300 < x ≤ 440 [Or Urine output < 500 mL/day] | x > 440 [Or Urine output < 200 mL/day] |

Note: Central Nervous System scoring algorithm has been included above for completeness but in Study 205821 it is not expected to form part of the overall SOFA total

In the SI.CONMEDS record (for vasopressors) the units may have to be converted from  $\mu g/min$  to  $\mu g/kg/min$  dose by merging on the weight from the vital signs dataset (and other unit conversions may be required for the other SOFA components).

PaO2/FiO2 values from the eCRF form should be double checked for accuracy (e.g. visual inspection of raw datasets to determine if they in the expected ranges for the stated unit).

#### 10.6.8. Oxygen Saturation

The oxygen saturation may be calculated from the provided ratio SaO2/FiO2 readout if the eCRF field for Oxygen Saturation (Vitals eCRF) is blank or missing.

#### 10.6.9. Calculation of PaO2 / FiO2 and SpO2 / FiO2

If required (e.g. because the automatically calculated eCRF field is blank or the units used in the auto-derived field appear to be incorrect) and sufficient source data are available then:

- The PaO2/FiO2 endpoint can be calculated when patients are intubated and have an arterial line present. Prior to computing the ratio the PaO2 may need to be converted from kPa units to mmHg using the conversion rate 1/0.133. FiO2 should be expressed as a proportion and not a percentage when deriving the ratio.
- SpO2/FiO2 will be calculated as a ratio of percentages.

#### 10.6.10. Construction of ARDATA.ALLCVTS

Guidance on the structure of the master A&R dataset that will hold potential covariate variables (for use in model building) is contained in Table 9.

Table 9 Suggested Metadata for ARADTA.ALLCVTS (Modifications may be made if required, e.g. to add/remove variables based on questions arising from observed data – the HARP metadata form would capture the final specification used). SAS label text and units to be added as appropriate to the data item.

| Type | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Info | STUDYID | STUDYID | ARDATA.CV (Unique list of subjid, centreid and visitnum |
| Info | SUBJID | SUBJID | combinations where at least one PASP and/or RV Size Ratio |
| Info | USUBJID | USUBJID | result was evaluable in CMANALFL=1 records) |
| Info | CENTREID | CENTREID | VISITNUM 20.00 = DAY 1 |
| Info | INVID | INVID | VISITNUM 30.00 = DAY 2 |
| Info | VISITNUM | VISITNUM | VISITNUM 40.00 = DAY 3 |
| Info | VISIT | VISIT | |
| Info | SUBJLEV | Extraction of set of subject level records | Only a single flag of 1 allowed per subject. Usually Day 1 record if present, day 2 (or 3) otherwise |
| Subject | AGE | Age at Screening | ARDATA.DEMO (AGE) |
| Subject | SEX | Sex | ARDATA.DEMO (SEX) |
| Subject | VSBMI | BMI at Screening | ARDATA.VITALS (VSBMI) |
| Subject | SAPSII | SAPS II at Screening | DMDATA.CC (Select CCORRSN where CCTESTCD=CC001) |
| Subject | RSINTU | Reason for Intubation at Screening (Categorical) | ARDATA.PR (Select the derived variable PRMIND which contains the mapping of the free text variable (PRINDC) for reason for intubation at screening visit (VISITNUM=10); see Section 10.6.4) |
| Time | INTUI | Intubated by Study Day (Binary Y/N) | ARDATA.PR (Where PRTREAT=INTUBATION & VISITNUM in (20,30,40)) For each subject and visitnum match: Set corresponding INTUI to Y if PROCCUR = Y for Day <i>; Set to N otherwise</i> |
| Subject | ARDSX | ARDS Diagnosis at any time (Binary Y/N) | DMDATA.FACE (Where FCETSTCD=FCEBU001) Set to Y if Any of FCEORSCD = ZZY for a subject; Set to N otherwise |

| Type | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Time | ARDSI | ARDS Diagnosis by Study Day (Binary | DMDATA.FACE (Where FCETSTCD=FCEBU001) |
| | | Y/N) | Treat any Screening results as being from Day 1 (use the worst |
| | | | case outcome as Day 1 result). For each subject and visitnum |
| | | | match: |
| | | | Set corresponding ARDSI to Y if FCEORSCD = ZZY for Day |
| | | | <i>; Set to N otherwise</i> |
| | | | Note: Class any SCREENING result as DAY 1 record for the |
| | | | purposes of ARDS diagnosis |
| Subject | INOX | Inhaled Nitric Oxide at any time (Binary | DMDATA.FACM (Where FCMTSTCD=FCMAX001) |
| | | Y/N) | Set to Y if Any of FCMORSCD = ZZY for a subject; Set to N |
| | 10101 | | otherwise |
| Time | INOI | Inhaled Nitric Oxide by Study Day (Binary | DMDATA.FACM (Where FCMTSTCD=FCMAX001) |
| | | Y/N) | Treat any Screening results as being from Day 1 (use the worst |
| | | | case outcome as Day 1 result). For each subject and visitnum |
| | | | match: |
| | | | Set corresponding INOI to Y if FCMORSCD = ZZY for Day <i>; Set to N otherwise</i> |
| Subject | VASOX | Vasopressor, Inotrope or other Vasoactive | DMDATA.FACM (Where FCMTSTCD=FCMAX002) |
| Subject | VASUA | agent at any time (Binary Y/N) | Set to Y if Any of FCMORSCD = ZZY for a subject; Set to N |
| | | agent at any time (binary 1714) | otherwise |
| Time | VASOI | Vasopressor, Inotrope or other Vasoactive | DMDATA.FACM (Where FCMTSTCD=FCMAX002) |
| 11110 | 77.001 | agent by Study Day (Binary Y/N) | Treat any Screening results as being from Day 1 (use the worst |
| | | agont 2) stady 2dy (2mary 1711) | case outcome as Day 1 result). For each subject and visitnum |
| | | | match: |
| | | | Set corresponding VASOI to Y if FCMORSCD = ZZY for Day |
| | | | <i>; Set to N otherwise</i> |
| Subject | PRONEX | Proned at any time (Binary Y/N) | ARDATA.PR (Where PRTREAT=MECHANICAL |
| • | | , | VENTILATION; exclude records with PRREFID=SOFA) |
| | | | Set to Y if Any of Subjects records have PRONE=Y |

| Туре | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Time | PRONEI | Proned by Study Day (Binary Y/N) | ARDATA.PR (Where PRTREAT=MECHANICAL VENTILATION |
| | | | & VISITNUM in (20,30,40); exclude records with |
| | | | PRREFID=SOFA) |
| | | | For each subject and visitnum match: |
| | | | Set corresponding PRONEI to Y if PRONE = Y for Day <i>; Set</i> |
| | | | to N otherwise |
| Subject | ECMOX | ECMO at any time (Binary Y/N) | ARDATA.PR (Where PRTREAT= EXTRACORPOREAL |
| • | | | MEMBRANE OXYGENATION) |
| | | | Set to Y if Any of Subjects records have PROCCUR=Y |
| Time | ECMOI | ECMO by Study Day (Binary Y/N) | ARDATA.PR (Where PRTREAT= EXTRACORPOREAL |
| | | | MEMBRANE OXYGENATION & VISITNUM in (20,30,40)) |
| | | | For each subject and visitnum match: |
| | | | Set corresponding ECMOI to Y if PROCCUR = Y for Day <i>;</i> |
| | | | Set to N otherwise |
| Subject | ECCO2RX | ECCO2R at any time (Binary Y/N) | ARDATA.PR (Where PRTREAT= EXTRACORPOREAL CO2 |
| - | | | REMOVAL) |
| | | | Set to Y if Any of Subjects records have PROCCUR=Y |
| Time | ECCO2RI | ECCO2R by Study Day (Binary Y/N) | ARDATA.PR (Where PRTREAT= EXTRACORPOREAL CO2 |
| | | | REMOVAL & VISITNUM in (20,30,40)) |
| | | | For each subject and visitnum match: |
| | | | Set corresponding ECCO2RI to Y if PROCCUR = Y for Day |
| | | | <i>; Set to N otherwise</i> |
| Subject | LCONDT | Last Contact Date (Date) | ARDATA.DS (Where DSSCATCD=4 & VISITNUM=0) |
| - | | | Select DSSTDT |
| Subject | LCONDY | Last Contact Study Day (Continuous) | ARDATA.DS (Where DSSCATCD=4 & VISITNUM=0) |
| • | | | Select DSSTDY |
| Subject | FUDT | Date of Follow Up Visit (Date) | DMDATA.VISIT (Where VISITNUM=50) |
| • | | . , , | Select VISITDT ` |

| Туре | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Subject | DTHHOSP | In hospital mortality (Categorical Y/N/U) | DMDATA.SS (Where VISITNUM=50 & SSTESTCD=AD009) |
| | | | Set to Y if SSORRSCD=ZZY; to N if SSORRSCD=ZZN and to |
| | | | U if SSORRSCD=ZZUNK |
| Subject | DERDTHDT | Derived Death Date (Date) | Set to the earliest of the dates obtained from |
| | | | DMDATA.DTH (match on SUBJID and select DDDT) |
| | | | Or |
| | | | LCONDT variable if DTHHOSP = Y |
| | | | Or |
| | | | If no dates located above but subject has DMDATA.STATUS |
| | | | DTHBWIND=Y then set to a derived date corresponding to day |
| | | | 3 (relative to that subjects date of 1st echo) |
| | | | Otherwise set to missing |
| Subject | DERDTHDY | Derived Death Study Day (Continuous) | The study day of the DERDTHDT (relative to time zero – the |
| | | | date of 1st echo) |
| | | | Set to missing if DERDTHDT = missing |
| Subject | DTH28 | Death by Day 28 (Categorical Y/N/U) | Set to Y if DERDTHDY not missing & ≤ 28 |
| | | | Set to N if [DERDTHDY = missing & LCONDY ≥ 28] or |
| | | | [DERDTHDY ≥ 28] |
| | | | Set to U otherwise |
| Subject | SURVIND | Survival Censoring Indicator (Categorical) | Set to 0 if DERDTHDT not missing |
| | | | Set to 1 (censored time) otherwise |
| | | | <note: be="" conjunction="" in="" indicator="" should="" td="" used="" variable="" with<=""></note:> |
| | | | LCONDY in any time to event analyses> |
| Subject | ICUDY | Length of stay (days) in ICU (Continuous) | DMDATA.HRU (Where HUCLVCD=4) |
| , | | | Select HUNDYCAR |
| Subject | HOSPDY | Length of stay (days) in Hospital | DMDATA.HRU (Where HUCLVCD=8) |
| - | | (Continuous) | Select HUNDYCAR |

| Type | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Subject | DYWOVNT | Ventilation Free Days (1 to 28) | DMDATA.HRU (Where HUSCATCD=3) |
| | | (Continuous) | Select DYWOVNT |
| Subject | SGX1TO3 | Any Surgery between Day 1 and Day 3 | DMDATA.SURGERY (Where VISITNUM=50) |
| | | (Binary Y/N) | Select SPYN |
| Time | RVDYSI | Single variable capturing RV Dysfunction | ARDATA.CV (Where CVANALFL=1 & CVTSTCD in (AK015, |
| | | Status by Study Day (Categorical: | AK016)) |
| | | 1=No PCD | For each subject and visitnum match Set to: |
| | | 2=Moderate PCD (not severe enough to | <ul> <li>1 if CVTSTCD=AK015 &amp; CVORRSCD=N</li> </ul> |
| | | qualify as ACP) | <ul> <li>2 if [CVTSTCD=AK015 &amp; CVORRSCD=Y] &amp;</li> </ul> |
| | | 3 = Non-severe ACP | [CVTSTCD=AK016 & CVORRSCD=51] |
| | | 4 = Severe ACP) | 3 if [CVTSTCD=AK015 & CVORRSCD=Y] & |
| | | | [CVTSTCD=AK016 & CVORRSCD=52] |
| | | | 4 if [CVTSTCD=AK015 & CVORRSCD=Y] & |
| | | | [CVTSTCD=AK016 & CVORRSCD=53] |
| Subject | RVDYSX | Single variable capturing Worst observed | MAX of RVDYSI variable (group by SUBJID) |
| , | | RV Dysfunction Status at any time | |
| | | (Categorical) | |
| Subject | PCDACPX | Any PCD or ACP at any time in study | Set to Y if RVDYSX in (2,3,4) |
| - | | (Binary Y/N) | Set to N otherwise |
| Time | PCDACPI | Any PCD or ACP by Study Day (Binary | Set to Y if RVDYSI in (2,3,4) |
| | | Y/N) | Set to N otherwise |
| Subject | NORVDYSX | Did not have PCD or ACP at any time in | Set to Y if RVDYSX = 1 |
| - | | study (Binary Y/N) | Set to N otherwise |
| Time | NORVDYSI | Did not have PCD or ACP on Study Day | Set to Y if RVDYSI = 1 |
| | | (Binary Y/N) | Set to N otherwise |
| Subject | PCDX | Worst case was PCD at any time in study | Set to Y if RVDYSX = 2 |
| | | (Binary Y/N) | Set to N otherwise |
| Time | PCDI | PCD on Study Day (Binary Y/N) | Set to Y if RVDYSI = 2 |
| | | | Set to N otherwise |

| Type | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Subject | ACPX | Worst case was ACP at any time in study | Set to Y if RVDYSX = 3 |
| | | (Binary Y/N) | Set to N otherwise |
| Time | ACPI | ACP on Study Day (Binary Y/N) | Set to Y if RVDYSI = 3 |
| | | | Set to N otherwise |
| Subject | SEVACPX | Worst case was Severe ACP at any time in | Set to Y if RVDYSX = 4 |
| | | study (Binary Y/N) | Set to N otherwise |
| Time | SEVACPI | Severe ACP on Study Day (Binary Y/N) | Set to Y if RVDYSI = 4 |
| | | | Set to N otherwise |
| Subject | ARDNOX | ARDS but no PCD or ACP at any time in | Set to Y if [ARDSX=Y & NORVDYSX=Y] |
| | | study (Binary Y/N) | Set to N otherwise |
| Subject | ARDPCDX | ARDS and worst case PCD at any time in | Set to Y if [ARDSX=Y & PCDX =Y] |
| | | study (Binary Y/N) | Set to N otherwise |
| Subject | ARDACPX | ARDS and worst case ACP at any time in | Set to Y if [ARDSX=Y & ACPX =Y] |
| | | study (Binary Y/N) | Set to N otherwise |
| Subject | ARDSACPX | ARDS and worst case Severe ACP at any | Set to Y if [ARDSX=Y & SEVACPX =Y] |
| | | time in study (Binary Y/N) | Set to N otherwise |
| Time | GII | Global Inhomogeneity Index (Continuous) | DMDATA.CC (Select CCORRSN where CCTESTCD=BY001 & |
| | | | VISITNUM in (20,30,40)) |

| Type | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Time | Variable Name <various signs="" vital=""> SYSBP DIABP HEART TEMP RESP VSPO2BLD VSMAP VSPPV</various> | Take names/properties directly from dataset (Continuous) | DMDATA.VITALS (Where VISITNUM in (20,30,40) & VSREFID ^= SOFA) Select (use same name) SYSBP DIABP HEART TEMP RESP VSPO2BLD VSMAP VSPPV |
| Time | OI | Oxygenation Index (Continuous) | Match on subjid and visitnum DMDATA.RE (Where VISITNUM in (20,30,40) & RETESTCD=AC002) Select REORRSN Match on subjid and visitnum |
| Time | PAO2 | Partial pressure of arterial O2 (mmHg) (Continuous) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID ^=SOFA & LBTESTCD=PAO2_BLP) For each subject select the most recent non-missing value from visitnum 10,20 (and set result to have visitnum=20) prior to merging by subject and visitnum Select LBORRESN |
| Time | PAO2DM | DateTime of PAO2 Sample (DateTime) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID ^=SOFA & LBTESTCD=PAO2_BLP) For each subject select the most recent non-missing LBORRESN value from visitnum 10,20 (and set result to have visitnum=20) prior to merging by subject and visitnum Combine LBDT and LBACTTM into a single datetime formatted variable |

| Type | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Time | PACO2 | Carbon dioxide partial pressure (mmHg) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID |
| | | (Continuous) | ^=SOFA & LBTESTCD=PCO2_BLP) |
| | | | For each subject select the most recent non-missing value from |
| | | | visitnum 10,20 (and set result to have visitnum=20) prior to |
| | | | merging by subject and visitnum |
| | | | Select LBORRESN |
| Time | LACT | Serum Lactate (mmol/L) (Continuous) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID ^=SOFA & LBTESTCD=LACT_PLC) |
| | | | For each subject select the most recent non-missing value from |
| | | | visitnum 10,20 (and set result to have visitnum=20) prior to |
| | | | merging by subject and visitnum |
| | | | Select LBORRESN |
| Time | HC03 | Serum Bicarbonate (mEq/L) (Continuous) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID |
| | | | ^=SOFA & LBTESTCD=HC03_PLC) |
| | | | For each subject select the most recent non-missing value from |
| | | | visitnum 10,20 (and set result to have visitnum=20) prior to |
| | | | merging by subject and visitnum |
| | | | Select LBORRESN |
| Time | PH | Blood pH (Continuous) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID |
| | | | ^=SOFA & LBTESTCD=PH_BLG) |
| | | | For each subject select the most recent non-missing value from |
| | | | visitnum 10,20 (and set result to have visitnum=20) prior to |
| | | | merging by subject and visitnum |
| | | | Select LBORRESN |
| Time | BASEXA | Base excess (arterial whole blood) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID |
| | | (mEq/L) (Continuous) | ^=SOFA & LBTESTCD=BASEXA_BLC) |
| | | | For each subject select the most recent non-missing value from |
| | | | visitnum 10,20 (and set result to have visitnum=20) prior to |
| | | | merging by subject and visitnum |
| | | | Select LBORRESN |

| Type | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Time | BDEFA | Base deficit (arterial whole blood) (mEq/L) (Continuous) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID ^=SOFA & LBTESTCD=BDEFA_BLC) For each subject select the most recent non-missing value from |
| | | | visitnum 10,20 (and set result to have visitnum=20) prior to merging by subject and visitnum Select LBORRESN |
| Time | TROPI | Troponin I (UG/L) (Continuous) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID ^=SOFA & LBTESTCD=TROPI_PLC) |
| | | | For each subject select the most recent non-missing value from visitnum 10,20 (and set result to have visitnum=20) prior to merging by subject and visitnum Select LBORRESN |
| Time | TROPT | Troponin T (UG/L) (Continuous) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID ^=SOFA & LBTESTCD=TROPT_PLC) For each subject select the most recent non-missing value from visitnum 10,20 (and set result to have visitnum=20) prior to merging by subject and visitnum Select LBORRESN |
| Time | PFSOFA | PaO2/FiO2 entered onto SOFA form (Continuous) | DMDATA.LAB (Where VISITNUM in (10,20,30,40) & LBREFID =SOFA & LBTESTCD=PAO2FI_BLQ) For each subject select the most recent non-missing value from visitnum 10,20 (and set result to have visitnum=20) prior to merging by subject and visitnum Select LBORRESN |
| Time | FIO2 | Fraction of Inspired Oxygen (%) (Continuous) | DMDATA.FAPR (Where VISITNUM in (20,30,40) & FPRTSTCD=FPRAW005) Select FPRORSN. Match on subjid and visitnum |

| Type | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Time | FIO2DM | DateTime of FIO2 Sample (DateTime) | DMDATA.FAPR (Where VISITNUM in (20,30,40) & FPRTSTCD=FPRAW005) Combine FPRDT and FPRTM into a single datetime formatted |
| | | | variable Match on subjid and visitnum |
| Time | PFDIFF | Difference between PaO2 and FiO2 | (PAO2DM - FIO2DM) converted into minutes |
| | | Sampling occasions (mins) | |
| Time | PFECRF | PaO2/FiO2 derived (Continuous) | PAO2 / (FIO2 / 100) |
| Time | PFECRF30 | PaO2/FiO2 (sampling within ±30 mins) (Continuous) | Select PFECRF if ABS(PFDIFF) $\leq$ 30; set to missing otherwise |
| Time | FPRBH001 | Static Respiratory System Compliance | DMDATA.FAPR (Where VISITNUM in (20,30,40) & |
| | | (mL/cm H2O) (Continuous) | FPRTSTCD= FPRBH001) |
| | | | Select FPRORSN. Match on subjid and visitnum |
| Time | FPRBH003 | Pressure Support Ventilation (Binary Y/N) | DMDATA.FAPR (Where VISITNUM in (20,30,40) & |
| | | | FPRTSTCD= FPRBH003) |
| | | | Match on subjid and visitnum |
| | | | Set Y if FPRORSCD=ZZY |
| | | | Set N otherwise |
| Time | FPRAB001 | Tidal Volume (mL) (Continuous) | DMDATA.FAPR (Where VISITNUM in (20,30,40) & |
| | | | FPRTSTCD= FPRAB001) |
| | | | Select FPRORSN. Match on subjid and visitnum |
| Time | FPRAB002 | Positive End Expiratory Pressure PEEP | DMDATA.FAPR (Where VISITNUM in (20,30,40) & |
| | | (cm H2O) (Continuous) | FPRTSTCD= FPRAB002) |
| | | | Select FPRORSN. Match on subjid and visitnum |
| Time | FPRAB003 | Peak Ventilatory Pressure (cm H2O) | DMDATA.FAPR (Where VISITNUM in (20,30,40) & |
| | | (Continuous) | FPRTSTCD= FPRAB003) |
| | | | Select FPRORSN. Match on subjid and visitnum |
| Time | FPRAB008 | Plateau Ventilatory Pressure (cm H2O) | DMDATA.FAPR (Where VISITNUM in (20,30,40) & |
| | | (Continuous) | FPRTSTCD= FPRAB008) |
| | | | Select FPRORSN. Match on subjid and visitnum |

| Type | Variable Name | Details | Suggestions for derivation / data source |
|---|---|---|---|
| Time | FPRBH004 | Mean Airway Pressure (cm H2O) | DMDATA.FAPR (Where VISITNUM in (20,30,40) & |
| | | (Continuous) | FPRTSTCD= FPRBH004) |
| | | | Select FPRORSN. Match on subjid and visitnum |
| Time | FPRBH005 | Driving Pressure (cm H2O) (Continuous) | DMDATA.FAPR (Where VISITNUM in (20,30,40) & |
| | | | FPRTSTCD= FPRBH005) |
| | | | Select FPRORSN. Match on subjid and visitnum |
| Time | <various and<="" echo="" endpoints="" td=""><td>Take from source dataset</td><td>ARDATA.STATSCAT (drop STUDYID, CENTREID, INVID,</td></various> | Take from source dataset | ARDATA.STATSCAT (drop STUDYID, CENTREID, INVID, |
| | the key RAS peptides> | | INVNAME, AGE, SEX, RACE, RACECD, ATRTCD, ATRTGRP, |
| | | | TRTCD, TRTGRP, USUBJID, VISIT, AH001AC, AK015, AK016 |
| | | | variables) |
| | | | Select remaining variables and match on subjid and visitnum |

# 10.7. Appendix 7: Reporting Standards for Missing Data

# 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as having completed the Day 3 assessments as shown in the SoA. |
| | Withdrawn subjects may be replaced in the study. |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures, unless<br/>otherwise specified (e.g. because they withdrew consent as detailed in the study<br/>protocol).</li> </ul> |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

# 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in participant listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| Missing<br>Categorical<br>Covariates | <ul> <li>In the statistical models of RAS peptides as predictors of measures of RV function (and other associated models), a number of categorical covariates (e.g. sex, prior history of RAS modulators, type of echocardiogram, use of vasopressors, proning status, use of nitric oxide) may be required. The following rules should be applied to variables that are to be included in the final statistical model:</li> <li>In the unlikely event that sex is not recorded for a participant, then data from that participant will not be included.</li> <li>For prior history of RAS modulators, a participant is assumed not to have had such a history unless explicitly reported otherwise.</li> <li>For the other variables listed above, which are recorded on each study day, the following imputation algorithm should be applied for missing values: <ul> <li>If the same variable is not missing on a previous study day (including screening, if applicable), impute the most recent known value.</li> <li>Otherwise, if the same variable is not missing on a subsequent study day, impute the value from the nearest time point after the missing one.</li> </ul> </li> <li>Otherwise, keep the value as missing and exclude the participant from the analysis</li> </ul> |

# 10.7.2.1. Handling of Missing and Partial Dates/Times

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be |

| Element | Reporting Detail |
|---|---|
| Events | recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: o Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events. Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used. Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.8. Appendix 8: Values of Potential Clinical Importance

#### 10.8.1. Laboratory Values

Note: Due to usage of local labs, care should be taken to ensure each supplied unit has been converted into the units given below before applying the PCI criteria (if applicable – any multipliers of LLN / ULN do not require units).

PCI values have been taken from Study ACE114622 (mild to moderate ARDS). Since no investigational product is being administered in this study any PCI flags will act more as an awareness for the study team when interpreting the RAS peptides / other clinical outcomes for those individuals. Any lab tests which the medical monitor has not specified PCI ranges for are denoted as "NA" but will still be reviewed as part of the Min/Max variables in the Summary tables.

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag<br>(Relative –<br>Multipliers of LLN) | High Flag<br>(Relative –<br>Multipliers of ULN) |
| Platelet Count | | | 0.4 | NA |
| Red Blood Cell (RBC) Count | | | NA | NA |
| While Blood Cell (WBC) Count (absolute) | | | 0.67 | 1.82 |
| Usemedahin | | Male | 0.67 | 1.03 |
| Haemoglobin | | Female | 0.67 | 1.13 |
| Hematocrit | Ratio of | Male | 0.3 | 0.54 |
| петнаюсті | 1 | Female | 0.3 | 0.54 |
| (Total) Neutrophils | | | NA | NA |
| Lymphocytes | | | NA | NA |
| Monocytes | | | NA | NA |
| Eosinophils | | | NA | NA |
| Basophils | | | NA | NA |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag<br>(Relative –<br>Multipliers of LLN) | High Flag<br>(Relative –<br>Multipliers of ULN) |
| Urea / BUN | | | NA | NA |
| Chloride | | | NA | NA |
| Creatinine | | | NA | 2 |
| Potassium | | | 0.86 | 1.10 |
| Sodium | | | NA | NA |
| Total CO <sub>2</sub> | | | NA | NA |
| Total Bilirubin | | | NA | NA |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag | High Flag |
| Troponin I<br>(Note: Has been spelt as<br>Troponon in Protocol) | ng/mL | | NA | > 0.04 |
| Troponin T<br>(Note: Has been spelt as<br>Troponon in Protocol) | ng/mL | | NA | > 0.10 |

# 10.8.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <85 | >160 |
| Diastolic Blood Pressure | mmHg | <45 | >100 |
| Heart Rate | bpm | <40 | >110 |

# 10.9. Appendix 9: Abbreviations & Trade Marks

# 10.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| BLQ | Below Limit of Quantification |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CPSR | Clinical Pharmacology Study Report (interchangeable with the CSR |
| | abbreviation) |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DIC | Deviance Information Criteria |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| LAR | Legally Acceptable Representative |
| LLN | Lower Limit of Normal |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |

| Abbreviation | Description |
|--------------|---------------------------------------------------------------|
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SoA | Schedule of Assessments (also known as Time and Events table) |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TBC | To Be Confirmed |
| TFL | Tables, Figures & Listings |
| ULN | Upper Limit of Normal |
| ULQ | Upper Limit of Quantification |

# 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |

## 10.10. Appendix 10: List of Data Displays

# 10.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|---|---|---|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Safety | 2.1 to 2.n | 2.1 to 2.n |
| Pharmacodynamic and / or Biomarker | 3.1 to 3.n | 3.1 to 3.n |
| Participant Status and / or Other Clinical Assessments | 4.1 to 4.n | 4.1 to 4.n |
| Statistical Modelling | 5.1 to 5.n | 5.1 to 5.n |
| Section | Listi | ngs |
| ICH Listings | 1 to | X |
| Other Listings | y to | ) Z |

#### 10.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|---|---|---|---|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Participant Status and / or Other Clinical Assessments | OCA_Fn | OCA_Tn | OCA_Ln |
| Statistical Modelling | SM_Fn | SM _Tn | SM _Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.10.3. Deliverables

| Delivery Priority <sup>1</sup> | Description |
|--------------------------------|-------------------------------------|
| SAC X | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 10.10.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title Programming Notes | | Deliverable<br>[Priority] |
| Subjec | Subject Disposition | | | | |
| 1.1. | Enrolled | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT, CONSORT | SAC 1 |
| 1.2. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC 1 |
| 1.3. | Safety | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | SAC 1 |
| Protoc | ol Deviations | | | | • |
| 1.4. | Safety | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC 1 |
| Popula | ation Analysed | | | | |
| 1.5. | Enrolled | SP1A | Summary of Study Populations | IDSL | SAC 1 |
| 1.6. | Enrolled | SP2A | Summary of Exclusions from the Safety/Evaluable/Completed/At Risk Populations | IDSL If possible separate page for each population (this may require non-standard wrapper macro to call the standard macro separately for each population) If the Evaluable with prohibited conmed population is different to evaluable add it in (otherwise footnote the evaluable table to indicate they are the same) | SAC 1 |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Demog | raphic and Bas | seline Characterist | tics | | |
| 1.7. | Safety | DM1 | Summary of Demographic Characteristics by PCD/ACP status | ICH E3, FDAAA, EudraCT Instead of the set of treatment variables (columns) please use "No PCD/ACP" and "Any PCD/ACP" and "All Participants" as columns to group the subjects As well as the standard set of demography items (Sex, Age, Age Group, Height, Weight, BMI) please also include the following Disease specific baseline variables (with units if applicable) to facilitate manuscript publication (mixture of continuous and categorical variables) Baseline should be the earliest non-missing value from SCREENING or DAY 1 visits. Do not display values from Days 2 or 3 (if multiple timepoints are available for an item) SAPSII, SOFA, PaO2/FiO2 (from SOFA form), PaO2, FiO2, PaCO2, Oxygenation Index, Reason for Intubation (use the mapped variable not free text results), Proned, Receiving Inhaled Nitric Oxide, "Managed with Vasopressors, inotropes or other vasoactive agents", ECMO, ECCO2R, Global Inhomogeneity Index, SpO2, Serum Lactate, Serum Bicarbonate, pH, Base excess (arterial whole blood), Base deficit (arterial whole blood), Central Venous Pressure, Static respiratory system compliance, Respiratory rate (not from vitals but from FAPR), Pressure support (Y/N), Tidal Volume, PEEP, Peak Pressure, Plateau Pressure, Mean Airway Pressure, Driving Pressure, In-hospital Mortality (Y/N/Unkown) Note: Summarise with n, Median, Lower and Upper quartiles, Min and Max: Length of stay in ICU, Length of stay in hospital, Ventilation free days | SAC 2 |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.8. | Safety | DM11 | Summary of Age Ranges | EudraCT | SAC 2 |
| Prior ar | Prior and Concomitant Medications | | | | |
| 1.9. | Safety | MH4 | Summary of Current Medical Conditions | ICH E3 | SAC 2 |
| 1.10. | Safety | MH4 | Summary of Past Medical Conditions | ICH E3 | SAC 2 |
| 1.11. | Safety | CM1 | Summary of Concomitant Medications | ICH E3 Exclude the SOFA related records | SAC 2 |
# 10.10.5. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serious | Adverse Even | nts | | | |
| 2.1. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT Conditional output: a listing on its own may be sufficient if there are few events. Display lines showing "Drug-related SAE" and "Drug-related Fatal SAE" should be omitted as there is no study drug involved. | SAC 2 |
| Labora | tory | | | | |
| 2.2. | Safety | LB1 | Summary of Clinical Chemistry Values by Timepoint | ICH E3 Exclude the SOFA related records There is no baseline in this study as there is no treatment being administered. Therefore the only data that can be presented is raw values rather than changes from baseline. | SAC 2 |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3. | Safety | LB1 | Summary of Haematology Values by Timepoint | ICH E3 Exclude the SOFA related records There is no baseline in this study as there is no treatment being administered. Therefore the only data that can be presented is raw values rather than changes from baseline. | SAC 2 |
| Vital Sig | gns | | | | |
| 2.4. | Safety | VS1 | Summary of Vital Signs by Timepoint | ICH E3 Exclude the SOFA related records There is no baseline in this study as there is no treatment being administered. Therefore the only data that can be presented is raw values rather than changes from baseline. | SAC 2 |

## 10.10.6. Pharmacodynamic and Biomarker Tables

| Pharma | codynamic an | d Biomarker: Tab | les | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Echoca | rdiography | | | | |
| 3.1. | Evaluable | PD_T1<br>(ECHO) | Summary of Echocardiogram Measurements by Timepoint | Two separate statistics tables: 1) for continuous, 2) for qualitative echo measurements. | SAC 1 |
| 3.2. | Evaluable | SM_T1<br>(ECHO) | Within- and Between-Subject Variability of Continuous Echocardiogram Measurements | | SAC 1 |
| RAS Bi | omarkers | | | | |
| 3.3. | Evaluable | PD_T2<br>(RAS) | Summary of RAS Biomarker Measurements by Timepoint | Present results for levels and log transformed in two separate tables. | SAC 1 |
| 3.4. | Evaluable | SM_T1<br>(RAS) | Within- and Between-Subject Variability of RAS Biomarker Measurements | | SAC 1 |

| Partic | Participant Status and Other Clinical Assessments: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Disea | Disease Diagnosis Status | | | | |
| 4.1. | At risk | OCA_T1<br>(DISEASE_INCIDENCE) | Summary of ARDS, PCD and ACP Incidence Rates by Timepoint and Study | Create two tables: 1) summarizing of number of the cases, where patient may contribute multiple times and 2) with overall incidence rates including the joint categories. Note: Shell does not contain all items to be displayed | SAC 1 |

# 10.10.7. Pharmacodynamic and Biomarker Figures

| Pharm | nacodynamic and | Biomarker: Figures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Echoo | ardiography | • | | | |
| 3.1. | Evaluable | PD_F2<br>(SCAT3D_YN) | Scatterplot of PASP vs RV Size Ratio marked by Paradoxical Septal Motion Status | Scatterplot of (x-axis) PASP vs (y-axis) RV size ratio. Paradoxical Septal Motion Status is marked by black(Y)-grey(N) colour. For Not Done PSM status leave blank (i.e. do not plot a coloured circle within the data point) | SAC 1 |
| RAS E | Biomarkers | | | | |
| 3.2. | Evaluable | PD_F1<br>(SCAT2D) | Scatterplots of Ang II, Ang(1-7) and Ang(1-5) combinations | Display with a Log10-transformed x and y axis scales. Separate page/plot for each combination. Present Ang II Vs Ang(1-7), Ang II Vs Ang(1-5) and Ang(1-7) Vs Ang(1-5) in | SAC 1 |
| 3.3. | Evaluable | PD_F4<br>(SERIES1D) | Individual Line Plots of RAS Biomarkers by Timepoint | On separate pages, time series plots for RAS biomarker readouts: Ang II, Ang(1-7), Ang(1-5), Ang II/Ang(1-7) ratio per visit (use log10 scale for yaxis). If the number of subject is too large omit the legend. | SAC 1 |

| Pharm | acodynamic and l | Biomarker: Figures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.4. | Evaluable | PD_F2<br>(SCAT3D_YN) | Scatterplots of Selected Echocardiography Endpoints Vs selected RAS biomarkers by Paradoxical Septal Motion Status | On separate pages, scatterplots of (x-axis) RAS biomarker readouts: Ang II, Ang(1-7), Ang(1-5), Ang II/ Ang(1-7) ratio (using log10 axis scale), vs (y-axis) PASP and RV size ratio readouts. Paradoxical Septal Motion Status is marked by black(Y)-grey(N) colour. For Not Done PSM status leave blank (i.e. do not plot a coloured circle within the data point) | SAC 1 |
| 3.5. | Evaluable | PD_F3<br>(SCAT3D_CONT) | Scatterplots of PASP vs. RV Size Ratio marked by RAS biomarker levels | On separate pages, scatterplots for (x-axis) PASP vs (Y-axis) RV size ratio coloured by RAS biomarker readouts: Ang II, Ang(1-7), ANG II/ Ang(1-7) ratio and Ang(1-5) on rainbow colour scale (no log-transformation). For each RAS biomarker scatterplot without and with visit marks provided. | SAC 1 |

## 10.10.8. Statistical Modelling Tables

| Statist | ical Modelling | : Tables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prepar | atory Analysis | 3 | | | |
| 5.1. | Evaluable | SM_T2<br>(BICORR_PHARM) | Bivariate Correlations of RAS Biomarkers with Pharmacodynamic Endpoints | Consider three different measures of correlation:1) derived from the bivariate mixed effect model and its between-marker Sigma vcov matrix 2) Pearson correlation 3) Spearman correlation A version of this output should be produced as soon as possible after the interim or final analysis has been triggered in order to enable the team to decide a) which covariates to include in the models and b) which of the conditional outputs (if any) to produce. List of continuous covariates to be provided at run time by statistician | SAC 1 |

| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 5.2. | Evaluable | SM_T2<br>(BICORR_CONT) | Bivariate Correlations of Ang II, Ang(1-7), PASP and RV Size Ratio with Continuous Covariates | Consider three different measures of correlation:1) derived from the bivariate mixed effect model and its between-marker Sigma vcov matrix 2) Pearson correlation 3) Spearman correlation A version of this output should be produced as soon as possible after the interim or final analysis has been triggered in order to enable the team to decide which covariates to include in the primary and secondary models. List of continuous covariates to be provided at run time by statistician | SAC 1 |
| 5.3. | Evaluable | SM_T3<br>(ECHO_RAS_<br>CAT) | Summary Statistics of RAS biomarkers and Echocardiogram<br>Endpoints by Categorical Covariates | A version of this output should be produced as soon as possible after the interim or final analysis has been triggered in order to enable the team to decide which covariates to include in the primary and secondary models. List of categorical covariates will be provided by statistician at time of analysis | SAC 1 |

| Statist | Statistical Modelling: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Statist | ical Modelling | | | | |
| 5.4. | Evaluable | SM_T4 (MODEL1) | Summary of Primary Model Results: Ang II as a Predictor of PASP and RV Size Ratio | On separate pages: Table 1) subtitle: Model Parameters Values with Statistics Table 2) subtitle: PASP and RV Model Predictions for Reference Ang II Values: Pre-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii _level=""> (pg/mL) Table 3) subtitle: Probability of RV Disfunction Given Reference Ang II Values: Pre-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii _level=""> (pg/mL) Add any sensitivity reference value results onto separate pages. For clear separation the subtitles start with 'SENSITIVITY:'</ang_ii></ang_ii_level></ang_ii></ang_ii_level> | SAC 1 |

| Statist | ical Modelling | : Tables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.5. | Evaluable | SM_T4 (MODEL2) | Summary of Secondary Model Results: Ang(1-7) as a Predictor of PASP and RV Size Ratio | On separate pages: Table 1) subtitle: Model Parameters Values with Statistics Table 2) subtitle: PASP and RV Model Predictions for Reference Ang(1-7) Values: Pre-dose < Ang(1-7)_level> (pg/mL) and Post-dose < Ang(1- 7)_level> (pg/mL) Table 3) subtitle: Probability of RV Disfunction Given Reference Ang(1-7) Values: Pre-dose < Ang(1-7)_level> (pg/mL) and Post-dose < Ang(1- 7)_level> (pg/mL) Add any sensitivity reference value results onto separate pages. For clear separation the subtitles start with 'SENSITIVITY:' | SAC 1 |

| Statist | Statistical Modelling: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.6. | Evaluable | SM_T4 (MODEL3) | Summary of Secondary Model Results: Ang(1-5) as a Predictor of PASP and RV Size Ratio | [conditional output] On separate pages: Table 1) subtitle: Model Parameters Values with Statistics Table 2) subtitle: PASP and RV Model Predictions for Reference Ang(1-5) Values: Pre-dose < Ang(1-5)_level> (pg/mL) and Post-dose < Ang(1- 5)_level> (pg/mL) Table 3) subtitle: Probability of RV Disfunction Given Reference Ang(1-5) Values: Pre-dose < Ang(1-5)_level> (pg/mL) and Post-dose < Ang(1- 5)_level> (pg/mL) Only analysis would be the sensitivity reference value, but still start the subtitles with 'SENSITIVITY:' | SAC 1 |
| 5.7. | Evaluable | SM_T4 (MODEL4) | Summary of Secondary Model Results: Ang II and Ang(1-7) as Joint Predictors of PASP and RV Size Ratio | [conditional output] Model only run if data permit | SAC 1 |

## 10.10.9. Statistical Modelling Figures

| Statist | Statistical Modelling: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Statist | ical Modelling | Figures | | | |
| 5.1. | Evaluable | SM_F1 | Scatterplot of PASP vs RV Size Ratio, Coloured by Ang II Value, with Posterior Prediction Regions for RV Function Measurements for Protocol-Defined Reference Values of Ang II | On separate pages: Figure 1) the scatterplot version with no visit marks and subtitle: Pre-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii_level> (pg/mL) Ang II Figure 2) the scatterplot version with visit marks and subtitle: Pre-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii_level> (pg/mL) Ang II Figure 3) subtitle: PASP Median and 95% Equal-Tailed Credibility Intervals for Pre-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii_level> (pg/mL) Ang II Figure 4) subtitle: RV size Median and 95% Equal-Tailed Credibility Intervals for Pre-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii_level> (pg/mL) Ang II Figure 5) subtitle: Prediction Regions for RV Function Measurements for Pre-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii_level> (pg/mL) and Post-dose <ang_ii_level> (pg/mL) Ang IIAdd any sensitivity reference value results onto separate pages. For clear separation the subtitles start</ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level></ang_ii_level> | SAC 1 |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| | | | | with 'SENSITIVITY:' | |
| 5.2. | Evaluable | SM_F1 | Scatterplot of PASP vs RV Size Ratio, Coloured by Ang(1-7) Value, with Posterior Prediction Regions for RV Function Measurements for Protocol-Defined Reference Values of Ang(1-7) | On separate pages: Figure 1) the scatterplot version with no visit marks and subtitle: Pre-dose <ang(1-7)_level> (pg/mL) and Post-dose <ang(1-7)_level> (pg/mL) Ang(1-7) Figure 2) the scatterplot version with visit marks and subtitle: Pre-dose <ang(1-7)_level> (pg/mL) and Post-dose <ang(1-7)_level> (pg/mL) and Post-dose <ang(1-7)_level> (pg/mL) Figure 3) subtitle: PASP Median and 95% Equal-Tailed Credibility Intervals for Pre-dose <ang(1-7)_level> (pg/mL) and Post-dose <ang(1-7)_level> (pg/mL) Ang(1-7) Figure 4) subtitle: RV size Median and 95% Equal-Tailed Credibility Intervals for Pre-dose <ang(1-7)_level> (pg/mL) and Post-dose <ang(1-7)_level> (pg/mL) and Post-dose <ang(1-7)_level> (pg/mL) and Post-dose <ang(1-7)_level> (pg/mL) Ang(1-7) Figure 5) subtitle: Prediction Regions</ang(1-7)_level></ang(1-7)_level></ang(1-7)_level></ang(1-7)_level></ang(1-7)_level></ang(1-7)_level></ang(1-7)_level></ang(1-7)_level></ang(1-7)_level></ang(1-7)_level></ang(1-7)_level> | SAC 1 |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| | | | | for RV Function Measurements for Pre-dose <ang(1-7)_level> (pg/mL) and Post-dose <ang(1-7)_level> (pg/mL) Ang(1-7) Add any sensitivity reference value results onto separate pages. For clear separation the subtitles start with 'SENSITIVITY:'</ang(1-7)_level></ang(1-7)_level> | |
| 5.3. | Evaluable | SM_F1 | Scatterplot of PASP vs RV Size Ratio, Coloured by Ang(1-5) Value, with Posterior Prediction Regions for RV Function Measurements for Protocol-Defined Reference Values of Ang(1-5) | [conditional output] On separate pages: Figure 1) the scatterplot version with no visit marks and subtitle: Pre-dose <ang(1-5)_level> (pg/mL) and Post-dose <ang(1-5)_level> (pg/mL) Ang(1-5) Figure 2) the scatterplot version with visit marks and subtitle: Pre-dose <ang(1-5)_level> (pg/mL) and Post-dose <ang(1-5)_level> (pg/mL) and Post-dose <ang(1-5)_level> (pg/mL) Ang(1-5) Figure 3) subtitle: PASP Median and 95% Equal-Tailed Credibility Intervals for Pre-dose <ang(1-5)_level> (pg/mL) Ang(1-5) Level&gt; (pg/mL) Ang(1-5) Figure 4) subtitle: RV size Median and 95% Equal-Tailed Credibility Intervals for Pre-dose <ang(1-5)_level> (pg/mL) and Post-dose <ang(1-5)_level> (pg/mL) and Post-dose <ang(1-5)_level> (pg/mL) Ang(1-5) Figure 5) subtitle: Prediction Regions</ang(1-5)_level></ang(1-5)_level></ang(1-5)_level></ang(1-5)_level></ang(1-5)_level></ang(1-5)_level></ang(1-5)_level></ang(1-5)_level></ang(1-5)_level> | SAC 1 |

| Statisti | Statistical Modelling: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | | for RV Function Measurements for<br>Pre-dose <ang(1-5)_level> (pg/mL)<br/>and Post-dose <ang(1-5)_level><br/>(pg/mL) Ang(1-5)<br/>Only analysis would be the sensitivity</ang(1-5)_level></ang(1-5)_level> | |
| | | | | reference value, but still start the subtitles with 'SENSITIVITY:' | |
| 5.4. | Evaluable | SM_F2 | Boxplots of Ang II, Ang(1-7), Ang(1-5), PASP and RV Size Ratio by Categorical Covariates. Auxiliary output for Table 5.3 | [conditional output] | SAC [1] |

## 10.10.10. ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | • | • |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC 1 |
| 2. | Enrolled | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC 1 |
| Protoc | ol Deviations | | | • | • |
| 3. | Safety | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC 1 |
| 4. | Enrolled | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC 1 |
| Popula | tions Analysed | | | • | • |
| 5. | Enrolled | SP3a | Listing of Subjects Excluded from Any Population | ICH E3 | SAC 1 |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 6. | Safety | DM2 | Listing of Demographic Characteristics | ICH E3 Use same set of variables as the corresponding summary table | SAC 2 |
| Prior a | nd Concomitan | t Medications | | | • |
| 7. | Safety | CP_CM3 | Listing of Concomitant Medications | IDSL<br>Exclude the SOFA related records | SAC 2 |
| Advers | e Events Section | on is not applicab | le as non-serious AEs are not being databased | | • |
| Seriou | s and Other Sig | nificant Adverse | Events | | |
| 8. | Safety | AE8CPa | Listing of Serious Adverse Events | ICH E3 | SAC 2 |
| 9. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC 2 |
| 10. | Safety | AECP8 | Listing of Serious Adverse Events Leading to Withdrawal from Study | ICH E3 | SAC 2 |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Lab | All Laboratory | | | | |
| 11. | Safety | LB5 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance | ICH E3 Exclude the SOFA related records | SAC 2 |
| Vital Sig | Vital Signs | | | | |
| 12. | Safety | VS4 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL<br>Exclude the SOFA related records | SAC 2 |

## 10.10.11. Non-ICH Listings

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acodynamic an | d Biomarker Listii | ngs | | |
| 13. | Evaluable | PD_L1 | Listing of Echocardiograph Measurements | Include all echo measures except the original eCRF PASP (AH001), AH001src, the programmatically derived variable containing the combined RAP (RAP), AK015 and AK016 which concern the ACP/PCD and its severity (those are displayed in Listing 19). Keep the order as in Section 5.5. Except for Estimated and Measured RAP have blank records if no result obtained for a test to maintain consistency of output for each subject and visit combination | SAC 1 |
| 14. | Evaluable | PD_L2 | Listing of RAS Biomarker Values | Listing on non-transformed levels. Include Ang II / Ang(1-7) ratio and ANG(1-5) | SAC 1 |
| Particip | oant Status and | Other Clinical As | sessments Listings | | |
| 15. | At Risk | OCA_L5 | Listing of Disease Diagnosis Status | Match to items in Table 4.1 | SAC 1 |
| 16. | Safety | AE2 (Modified) | Listing of Relationship between Reasons for Intubations and Verbatim Text | Display the Mapped categories (in place of System Organ Class – in the order implied in Section 10.6.4) and all of the free text reasons within each mapping (in place of Verbatim text) and omit the Preferred Term column (from the AE2 shell) | SAC 1 |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Statisti | cal Modelling L | istings | | | |
| 17. | Evaluable | SM_L1 | Listing of Primary Statistical Model Output: Ang II as a Predictor of PASP and RV Size Ratio | Start with Gelman-Rubin diagnostics for model parameters convergence given different starting points. Mark considered burn-in period. Further, include model printouts from PROC MCMC for parameter estimates and PASP and RV Size Ratio predictions given Ang II reference values. | SAC 1 |
| 18. | Evaluable | SM_L1 | Listing of Secondary Model Results: Ang(1-7) as a Predictor of PASP and RV Size Ratio | Start with Gelman-Rubin diagnostics for model parameters convergence given different starting points. Mark considered burn-in period. Further include model printouts from PROC MCMC for parameter estimates and PASP and RV Size Ratio predictions given Ang(1-7) reference values. | SAC 1 |
| 19. | Evaluable | SM_L1 | Listing of Secondary Model Results: Ang(1-5) as a Predictor of PASP and RV Size Ratio | [conditional output] Start with Gelman-Rubin diagnostics for model parameters convergence given different starting points. Mark considered burn-in period. Further include model printouts from PROC MCMC for parameter estimates and PASP and RV Size Ratio predictions given Ang(1-5) reference values. | SAC 1 |
| 20. | Evaluable | SM_L1<br>(Modified for<br>model structure<br>/ parameters) | Listing of Secondary Model Results: Ang II and Ang(1-7) as Joint Predictors of PASP and RV Size Ratio | [conditional output] | SAC 1 |

## 10.11. Appendix 11: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request